# A <u>Pragmatic Randomized trial Evaluating Pre-operative</u> <u>Alcohol skin solutions in <u>FRactured Extremities</u> (PREPARE Closed): Statistical Analysis Plan</u>

**Trial Registration:** clinicaltrials.gov, NCT03523962. Registered May 14, 2018, https://clinicaltrials.gov/ct2/show/NCT03523962

**SAP Version:** 1.0

**Protocol Version: 2.2** 

**SAP Revisions:** None

**Disclaimer:** This SAP was adapted from the Aqueous-PREP (Aqueous skin antisepsis before surgical fixation of open fractures) SAP, which was published in *Trials* in September 2022 (https://trialsjournal.biomedcentral.com/articles/10.1186/s13063-022-06541-0). A copy of the Aqueous-PREP SAP was also uploaded onto the ClinicalTrials.gov trial registration page (https://clinicaltrials.gov/ct2/show/NCT03385304). The Aqueous-PREP primary manuscript was published in *The Lancet* in October 2022 (https://www.thelancet.com/journals/lancet/article/PIIS0140-6736(22)01652-X/fulltext#seccestitle200).

| Reviewed and Approved by: | | |
|---|---|---|
| Dr. Gerard Slobogean<br>(Principal Investigator) | Signature: 61 evard Slobogean 7DFE42965445427 | Date: 22-Feb-2023 |
| Dr. Sheila Sprague<br>(Principal Investigator) | Signature: Docusigned by: Inula - Sprague OEB2EE3A208BA52 | Date: 21-Feb-2023 |
| Dr. Nathan N. O'Hara<br>(Statistician) | Signature: Docusigned by: Nathan O'Hara | Date: 21-Feb-2023 |
| Diane Heels-Ansdell<br>(Statistician) | Signature: A15DD93C7A70439 Docusigned by: | Date: 27-Feb-2023 |
| Sofia Bzovsky<br>(Statistical Analyst) | Signature: CAA2CFEEFA2342A Sofia Booksky | Date: 21-Feb-2023 |

#### **ABSTRACT**

## **Background**

Approximately 5% of closed fractures that are treated operatively will develop a surgical site infection. The PREPARE Closed trial will investigate the effect of iodine povacrylex (0.7% free iodine) in 74% isopropyl alcohol versus 2% chlorhexidine gluconate in 70% isopropyl alcohol antiseptic solutions in reducing infections after surgery for closed lower extremity or pelvic fractures. The study protocol was published in April 2020.

#### **Methods and Design**

The PREPARE Closed trial is a pragmatic, multicentre, open-label, randomized multiple period cluster crossover trial. Each participating cluster is randomly assigned in a 1:1 ratio to provide 1 of the 2 study interventions on all eligible patients during a study period. The intervention periods are 2 months in length. After completing a 2-month period, the participating cluster crosses over to the alternative intervention. We plan to enroll a minimum of 6280 patients at 23 sites.

#### Results

The primary outcome is surgical site infection guided by the Centers for Disease Control and Prevention's National Healthcare Safety Network reporting criteria (2017). All participants' surgical site infection surveillance period will end 30 days after definitive fracture management surgery for superficial infections and 90 days after definitive fracture management surgery for deep incisional or organ/space infections. The secondary outcome is an unplanned fracture-related reoperation within 12 months of the fracture.

## Conclusion

This manuscript serves as the formal statistical analysis plan (version 1.0) for the PREPARE Closed trial. The statistical analysis plan was completed on February 21, 2023.

# Keywords

Closed fracture, surgical site infection, alcohol antiseptic solutions

#### 1.0 INTRODUCTION

## 1.1 Background and Rationale

The prevention of infection is a critical goal of perioperative care for patients with surgically treated fractures of the closed lower extremity or pelvis. Surgical site infections are often devastating complications because of the unplanned reoperations, fracture healing difficulties, and adverse events from prolonged antibiotic treatments. Ultimately, infectious complications in these fracture populations lead to prolonged morbidity, loss of function, and potential limb loss.

Standard practice in the management of extremity fractures includes cleaning the injured limb with an antiseptic skin solution in the operating room prior to making a surgical incision. The available solutions kill bacteria and decrease the quantity of native skin flora, thereby reducing surgical site infection.<sup>2–5</sup> While there is extensive guidance on specific procedures for prophylactic antibiotic use and standards for sterile technique, the evidence regarding the choice of antiseptic skin preparation solution is very limited for extremity fracture surgery.

The PREPARE Closed trial will provide the necessary evidence to guide the choice of antiseptic skin solution to prevent surgical site infections in patients with closed lower extremity or pelvic fractures. The trial is poised to significantly impact the care and outcomes of closed lower extremity or pelvic fracture patients.

#### 1.2 Objectives

The overall objective of the PREPARE Closed trial is to compare the effect of iodine povacrylex (0.7% free iodine) in 74% isopropyl alcohol versus 2% chlorhexidine gluconate in 70% isopropyl

alcohol antiseptic solutions for the surgical management of closed lower extremity or pelvic fractures.

Primary Objective and Hypothesis

To determine the effect of iodine povacrylex (0.7% free iodine) in 74% isopropyl alcohol versus 2% chlorhexidine gluconate in 70% isopropyl alcohol antiseptic solutions in preventing surgical site infections. We hypothesize that iodine povacrylex in alcohol antiseptic will be more effective in preventing surgical site infections than chlorhexidine gluconate in alcohol antiseptic.<sup>5,6</sup>

Secondary Objective and Hypothesis

To determine the effect of iodine povacrylex (0.7% free iodine) in 74% isopropyl alcohol versus 2% chlorhexidine gluconate in 70% isopropyl alcohol antiseptic solutions in preventing unplanned fracture-related reoperations. We hypothesize that iodine povacrylex in alcohol antiseptic will be more effective in preventing unplanned reoperations than chlorhexidine gluconate in alcohol antiseptic.<sup>5,6</sup>

Subgroup Objectives and Hypotheses

We will perform two subgroup analyses to determine if the effects of preoperative antiseptic skin solutions on surgical site infection vary within clinically relevant subgroups. The subgroups will be defined by i) the presence or absence of the soft tissue injury (defined as severe soft tissue injury versus no severe soft tissue injury); and ii) the presence or absence of a periarticular fracture. We hypothesize that the magnitude of the effect of iodine povacrylex (0.7% free iodine) in 74% isopropyl alcohol compared with 2% chlorhexidine gluconate in 70% isopropyl alcohol antiseptic

in preventing surgical site infections will be greater in severe soft tissue injuries and in the presence of periarticular fractures.

## 1.3 Reporting

The structure of this statistical analysis plan follows the Guidelines for the Content of Statistical Analysis Plans in Clinical Trials.<sup>7</sup> The reporting of the trial results will follow the 2010 CONSORT statement and the extension statements for Cluster Trials and Randomized Crossover Trials, as applicable.<sup>8</sup> Additional statistical analyses plans will be developed for secondary analyses of the trial data.

#### 2.0 STUDY METHODS

## 2.1 Trial Design

1

2

9

10

17

18

- 3 The study is a pragmatic, multicentre, open-label, randomized multiple period cluster crossover
- 4 trial. We defined clusters as orthopaedic practices within participating hospitals, with each
- 5 participating hospital having only one participating orthopaedic practice. <sup>9</sup> The intervention periods
- 6 are approximately 2 months in length. After completing a 2-month period, the participating cluster
- 7 crosses over to the alternative intervention where they use the other study solution for the next 2-
- 8 month period. There are no washout periods between treatment periods.

#### 2.2 Randomization

- 11 The order of treatment allocation for each orthopaedic practice (cluster) will be randomly assigned
- using a computer-generated randomization table. Each cluster will start with the initially allocated
- study solution and crossover to the other solution for their second recruitment period. This process
- of alternating treatments will repeat approximately every 2 months as dictated by the initial
- 15 randomization until enrollment targets are met. The randomization will be in a 1:1 ratio,
- unrestricted, and executed only prior to the first sequence.

## 2.3 Sample Size

- 19 A sample size of 6280 patients will have 80% power to detect a 36% reduction in the odds of
- 20 infection with a two-sided alpha of 0.05. This estimate allows for a 10% loss to follow-up and
- assumes a baseline infection risk of 3.5%, 10 recruiting clusters, no between-period variance, and
- a 0.095 between-cluster variance. After the initial power calculations, we determined that
- 23 additional clusters were required to meet the study timelines. As such, we increased the number of

24 clusters from 10 to a minimum of 23. The increase in clusters results in a marginal increase in 25 statistical power (approximately 2%). 26 27 2.4 Framework 28 All study outcomes will be tested for superiority. 29 30 2.5 Interim Analysis and Stopping Guidance 31 PREPARE Closed does not have a planned interim analysis. However, the trial's Data and Safety 32 Monitoring Committee reviews the reporting of serious adverse events biannually and can 33 recommend early stopping if safety concerns are identified. 34 35 2.6 Timing of Outcome Assessments 36 Research personnel will contact study participants at 6 weeks, 3 months, 6 months, 9 months, and 37 12 months after their fracture. Our primary outcome will be surgical site infection (SSI) and it will 38 be assessed at 30 days (superficial infections) and at 90 days (deep and organ space infections) 39 after definitive fracture management surgery. The secondary outcome will be occurrence of an 40 unplanned fracture-related reoperation within 12 months of the fracture. Additional time points 41 will be used for our planned sensitivity analyses. 42 43 44

46

48

49

50

51

52

53

55

56

57

58

59

60

61

62

63

64

65

66

67

#### 3.0 STATISTICAL PRINCIPLES

3.1 Confidence Intervals and P-Values

47 All statistical tests will be two-sided and performed using a 5% significance level. We will report

all confidence intervals as 95% and two-sided. All results will be expressed as odds ratios produced

by analyses described in section 5.2. Interaction p-values will be provided for the subgroup

analyses. We will not adjust for multiple testing, and all sensitivity analyses and secondary results

will be interpreted as exploratory.

#### 3.2 Adherence and Protocol Deviations

Adherence will be assessed at the definitive fracture surgery for each participant and will be binary

in its definition. We will report adherence as the number and percentage of participants who

received the allocated intervention at their definitive fracture management surgery. If the

participant has multiple closed fractures and received the non-allocated treatment at the definitive

fracture management surgery for any of their closed fractures, we will consider them non-adherent.

We will also tabulate the reasons for non-adherence. The adherence percentages and reasons for

non-adherence will be reported by treatment arm.

Our rationale for defining adherence based solely on the antiseptic solution used during the

definitive fracture management surgery is that the vast majority of closed fractures do not require

staged surgical management and that the definitive fracture management surgery involves the final

implantation of the surgical fixation hardware, when it is most susceptible to bacterial

contamination and biofilm development.

3.3 Analysis Populations

Intention-to-Treat: Our primary analysis will use the intention-to-treat approach and will include all enrolled patients in the treatment groups to which their cluster was allocated at the time of their first fracture management surgery.

As-Treated: One of our sensitivity analyses will be performed on an as-treated population (see Section 5.4). The as-treated population will include participants from the intention-to-treat population but classified based on the intervention received at their definitive fracture management surgery. Participants who do not receive one of the two study interventions will be excluded from this analysis. This approach for defining the as-treated treatment groups is a simpler adaptation of what was initially proposed in the protocol. This final approach was selected to be consistent with the classification of adherence outlined above.

#### 4.0 TRIAL POPULATION

## 4.1 Cluster Screening and Eligibility

Prior to commencing the trial, the investigators solicited orthopaedic surgery practices treating patients with closed fracture(s) of the lower extremity or pelvis in hospitals in the United States and Canada to participate in the trial. All potential clusters completed a feasibility questionnaire prior to initiating start-up activities. To be included in the trial, each cluster had to demonstrate: 1) adequate research personnel infrastructure to manage the study, 2) adequate fracture patient volume to complete enrolment within the study timeline, 3) a commitment from all surgeons to adhere to the assigned interventions, and 4) the ability to procure both study interventions. All hospitals started with a run-in phase of at least 1 month to demonstrate that they could adhere to the trial protocol prior to commencing the study.

We will report the number of clusters (orthopaedic practices) screened, included, and excluded in a flow diagram. The number of clusters excluded by reason has been reported previously. Cluster randomization allocation will be included in the flow diagram, and adherence with treatment allocation during the run-in period by cluster will be summarized using percentages.

## 4.2 Patient Screening and Eligibility

All patients 18 years of age or older who present to a recruiting hospital for treatment of a closed fracture(s) of the lower extremity or pelvis will be screened by a research staff member for participation within 6 weeks of their fracture. Eligible patients must receive surgical incision (i.e., for fracture reduction or implant insertion), and the closed fracture(s) must be managed definitively with a surgical implant (e.g., internal fixation, external fixation, joint prosthesis, etc.). Written

informed consent is required for study enrollment to permit the clinical follow-up of study participants. However, our institutional review board did not require informed consent to occur prior to the study treatment, given the urgent nature of the surgery and the predetermination of the two commonly used interventions with cluster-crossover design. The patients, treating clinicians, and research team members at the participating sites are unmasked to the treatment allocation.

The number of patients screened, included, and excluded will be presented in a flow diagram (**Figure 1**). The figure will consist of the number of patients who were eligible, ineligible, and enrolled. In addition, the number of patients excluded by reason will be summarized. We will also list the number of participants who were enrolled and subsequently deemed ineligible by the Central Adjudication Committee by treatment group and overall. Participants deemed ineligible by a central adjudication committee blinded to the treatment will not be included in any analysis, as per the guidance of Fergusson et al.<sup>10</sup>

## 4.3 Participant Withdrawal

The level of withdrawal will be tabulated and classified as "withdrawal of consent" or "lost to follow-up". Participant deaths will also be tabulated.

#### 4.4 Participant Follow-Up

We will report the number of participants who complete follow-up at 3 months after definitive fracture management surgery and 12 months after their fracture, stratified by treatment allocation.

#### 4.5 Cluster Characteristics

Specific details on characteristics of participating clusters, orthopaedic characteristics, and surgical infection prevention information in the PREPARE Closed trial have been previously published.<sup>9</sup>

131

132

133

134

135

136

137

138

139

140

141

142

143

144

145

146

147

148

128

129

130

### 4.6 Participant Demographics, Fracture Characteristics, and Descriptions of Surgical and

#### **Perioperative Care**

We will describe the study population with respect to age, sex, race or ethnicity, body mass index, diabetes status, smoking status, Injury Severity Score, the American Society of Anesthesiologists Physical Status Classification System, the number of included closed fractures per participant, the presence of a severe soft tissue injury (defined as severe soft tissue injury versus no severe soft tissue injury), 11 the location of the fracture, the use of temporary fracture stabilization, number of planned surgeries, the duration of perioperative antibiotic administration, and the method of wound closure (Tables 1 and 2). Categorical data will be summarised by counts with percentages. Age will be summarised as a mean with standard deviation. We will report the Injury Severity Score as a median with an interquartile range. The duration of systemic perioperative antibiotics will be summarised in days and reported as a median with interquartile range. Body mass index (BMI) will be reported in kg/m<sup>2</sup> and subcategorized as underweight (BMI < 18.5), normal weight (18.5 -24.9), overweight (25 -29.9), and obese (BMI > 30). Additional patient characteristics may be reported as supplemental information. All reporting will be stratified by treatment groups. We will not statistically test for differences in baseline characteristics between treatment groups; however, the clinical importance of any imbalance will be noted.

#### 5.0 ANALYSIS

#### **5.1 Outcome Definitions**

151 Primary Outcome

Our primary outcome is SSI guided by the Centers for Disease Control and Prevention's (CDC) National Healthcare Safety Network reporting criteria (2017). The SSI surveillance period for all participants, including participants with multiple planned fracture surgeries, will end 30 days after definitive fracture management surgery for superficial SSI and 90 days after definitive fracture management surgery for deep incisional or organ/space SSI. We will also separately report but not statistically test the occurrence of each type of SSI (superficial incisional infections by 30 days, deep incisional infections by 90 days, and organ/space infections by 90 days) by treatment arm. If multiple tissue levels are involved in the infection, the type of SSI will be defined by the deepest tissue layer involved during the surveillance period. Therefore, only one type of SSI per participant will be reported.

CDC National Healthcare Safety Network Surgical Site Infection Reporting Criteria (2017)

| Outcome | Description |
|---|---|
| Superficial | Date of event for infection may occur from the date of fracture to 30 days after the definitive |
| Incisional | fracture management surgery |
| SSI | AND |
| | involves only skin and subcutaneous tissue of the incision |
| | AND |
| | patient has at least one of the following: |
| | a. purulent drainage from the superficial incision. |
| | b. organisms identified from an aseptically obtained specimen from the superficial |
| | incision or subcutaneous tissue by a culture or non-culture based microbiologic |
| | testing method which is performed for purposes of clinical diagnosis or |
| | treatment (e.g., not Active Surveillance Culture/Testing [ASC/AST]). |
| | c. superficial incision that is deliberately opened by a surgeon, attending physician |
| | or other designee and culture or non-culture-based testing is not performed. |
| | AND |
| | patient has at least one of the following signs or symptoms: pain or tenderness; |
| | localized swelling; erythema; or heat. |
| | <ul> <li>d. diagnosis of a superficial incisional SSI by the surgeon or attending physician<br/>or other designee.</li> </ul> |
| | The following do not qualify as criteria for meeting the definition of superficial SSI: |
| | Diagnosis/treatment of cellulitis (redness/warmth/swelling), by itself, does not meet |
| | \ |
| | criterion "d" for superficial incisional SSI. Conversely, an incision that is draining or that |

| Outcome | Description |
|---|---|
| | has organisms identified by culture or non-culture-based testing is not considered a |
| | cellulitis. |
| | A stitch abscess alone (minimal inflammation and discharge confined to the points of |
| | suture penetration). |
| | • A localized stab wound or pin site infection. Such an infection might be considered either |
| | a skin (SKIN) or soft tissue (ST) infection, depending on its depth, but not an SSI<br>Note: A laparoscopic trocar site for an operative procedure is not considered a stab wound. |
| | An infected burn wound is classified as BURN and is not an SSI. |
| Deep | The date of event for infection may occur from the date of fracture to 90 days after the definitive |
| Incisional | fracture management surgery |
| SSI | AND |
| | involves deep soft tissues of the incision (e.g., fascial and muscle layers) |
| | AND |
| | patient has at least one of the following: |
| | a. purulent drainage from the deep incision. |
| | b. a deep incision that spontaneously dehisces, or is deliberately opened or aspirated by a |
| | surgeon, attending physician or other designee, and organism is identified by a culture or non-culture based microbiologic testing method which is performed for purposes of |
| | clinical diagnosis or treatment (e.g., not Active Surveillance Culture/Testing |
| | [ASC/AST]) or culture or non-culture based microbiologic testing method is not |
| | performed |
| | AND |
| | patient has at least one of the following signs or symptoms: fever (>38°C); localized |
| | pain or tenderness. A culture or non-culture-based test that has a negative finding does |
| | not meet this criterion. |
| | c. an abscess or other evidence of infection involving the deep incision that is detected on |
| Organ/Space | gross anatomical or histopathologic exam, or imaging test Date of event for infection may occur from the date of fracture to 90 days after the definitive |
| SSI | fracture management surgery |
| 551 | AND |
| | infection involves any part of the body deeper than the fascial/muscle layers, that is opened or |
| | manipulated during the operative procedure |
| | AND |
| | patient has at least one of the following: |
| | a. purulent drainage from a drain that is placed into the organ/space (e.g., closed |
| | suction drainage system, open drain, T-tube drain, CT guided drainage) |
| | b. organisms are identified from an aseptically obtained fluid or tissue in the organ/space by a culture or non-culture based microbiologic testing method |
| | which is performed for purposes of clinical diagnosis or treatment (e.g., not |
| | Active Surveillance Culture/Testing [ASC/AST]). |
| | c. an abscess or other evidence of infection involving the organ/space that is |
| | detected on gross anatomical or histopathologic exam, or imaging test evidence |
| | suggestive of infection. |
| | AND |
| | meets at least one criterion for a specific organ/space infection site summarized in the |
| test and i | Surveillance Definitions for Specific Types of Infections chapter. <sup>1</sup> |

<sup>\*</sup>The CDC criteria have been modified to include all definitive fracture management surgeries instead of including only National Healthcare Safety Network procedures that require infection reporting.

## Secondary Outcome

The secondary outcome is the occurrence of an unplanned fracture-related reoperation within 12 months of the fracture. Unplanned reoperations are a common, patient-important outcome in fracture surgery research that captures severe wound and bone healing complications that may be related to occult infections. <sup>12–14</sup> Our definition includes treatments for infection, wound healing complications, or fracture healing complications such as a delayed union or nonunion. We will also report the occurrence of each type of unplanned reoperation by treatment arm.

# **5.2** Analysis Methods

We will report the number and percentage of patients who sustain the study outcomes by treatment group. We will evaluate the effect of the preoperative antiseptic solutions on our study outcomes using mixed effects regression models with a binomial distribution to produce treatment effect estimates presented as odds ratios with 95% confidence intervals as recommended. For patients with multiple closed fractures, the patient will remain the unit of analysis regardless of whether the study event occurs in one or more of their closed fractures. As suggested by Morgan et al. and Hemming et al., we will include time and treatment as fixed effects and use random effects to account for the complex correlation structure. We will consider three correlation structures, in the following sequence: exponential decay, nested exchangeable, and exchangeable. If we experience convergence issues or find insufficient between-period correlation to support an exponential decay or nested exchangeable structure, we will assume an exchangeable correlation structure. If we encounter convergence issues even with this model, a more simplified structure will be considered. The models will also include prespecified covariates prognostic of infection or unplanned reoperation as fixed effects, which includes the presence or absence of a severe soft

tissue injury and the presence or absence of a periarticular fracture.<sup>19</sup> The same covariates will be used for all primary and secondary outcomes. This planned analysis is a more complex structure than we proposed in the initial study protocol but represents the most recently recommended statistical techniques for cluster-crossover trial analysis.<sup>16,18,20,21</sup> Estimated within-period intracluster correlation coefficients will also be reported.<sup>22</sup>

Our primary and secondary analyses will use multiple imputations to account for missing data. The multiple imputation analysis will create 100 imputed datasets using multivariate imputation by chained equations and pooled using Rubin's rules for combining.<sup>23</sup> The imputation will be

## 5.3 Subgroup Analyses

performed separately within each treatment arm.

To determine treatment effect heterogeneity on the study outcomes, we will use the same analytical approach as specified for the primary and secondary outcomes above but include a treatment by subgroup interaction term in the model. We will report results by the prespecified subgroups, which consists of the presence or absence of a severe soft tissue injury (defined as severe soft tissue injury versus no severe soft tissue injury) and the presence or absence of a periarticular fracture (defined as AO/OTA fracture types 33, 41, 43 and 44 versus all other included fractures). The results of the subgroup analyses will be reported using a forest plot reporting odds ratios with 95% confidence intervals. These analyses will be approached and reported in accordance with best practices and guidelines for subgroup analyses. We will use the criteria suggested by Schandelmaier et al. to guide inferences about the credibility of our subgroup analyses. As participants may have more than one included fracture representing different subgroups, the

216

217

218

219

220

221

222

223

224

225

226

227

228

229

230

231

232

233

234

235

236

237

analyses will be performed by categorizing participants according to the fracture with the most severe injury characteristic for each subgroup. **5.4 Sensitivity Analyses** We will consider four alternative analysis approaches to evaluate the robustness of our findings, including alternative definitions of the primary outcome, an as-treated analysis of the primary and secondary outcomes, a complete case missing data analysis of the primary and secondary outcomes, and a Bayesian analysis of the primary and secondary outcomes. We will also allow for post-hoc sensitivity analysis based on information not anticipated in advance. Alternative Definitions of SSI: To evaluate the robustness of the result, we will consider two alternative exploratory definitions of SSI: 1) using the confirmatory criteria from the consensus definition of Fracture-Related Infection (FRI), and 2) expanding the CDC criteria for all types of SSI to within 1 year of injury.<sup>29</sup> Our adjudication of Fracture-Related Infection is defined by the confirmatory criteria outlined in its 2018 consensus definition.<sup>29</sup> The FRI criteria have been selected as an exploratory outcome because the CDC criteria have been criticized for failing to adequately account for the complexities of infections in traumatic fractures. 30,31 The FRI criteria attempt to improve the ability to detect infections specifically in fracture patients; however, this definition of FRI has not been fully validated or widely adopted. The confirmatory criteria include the presence of one or more of the following signs/symptoms:

- 238 1) Fistula, sinus, or wound breakdown (with communication to the bone or the implant).
  - 2) Purulent drainage from the wound or presence of pus during surgery.
    - 3) Phenotypically indistinguishable pathogens identified by culture from at least two separate deep tissue/implant (including sonication-fluid) specimens taken during an operative intervention. In the case of tissue, multiple specimens (3) should be taken, each with clean instruments (not superficial or sinus tract swabs). In cases of joint effusion arising in a joint adjacent to a fractured bone, fluid samples obtained by sterile puncture may be included as a single sample.
    - 4) Presence of microorganisms in deep tissue taken during an operative intervention, as confirmed by histopathological examination using specific staining techniques for bacteria or fungi.

The second exploratory definition of surgical site infection expands the CDC criteria to a 12-month surveillance period. This outcome will use the same diagnostic CDC reporting criteria for the primary; however, the timeframe for this outcome will be expanded to include all SSIs that occur within 12 months of fracture. Similar to the rationale for using the FRI outcome and the recommendations for a minimum of 12 months follow-up for orthopaedic fracture outcomes, this expanded timeframe will detect infections that occur beyond the standard CDC surveillance reporting periods. This modification of the CDC reporting periods has been used in previous orthopaedic fracture trials. 12,32

As-Treated Analysis: One of our sensitivity analyses will be performed on an as-treated population.

The as-treated population will include participants from the intention-to-treat population who

received one of the two interventions; however, participants will be classified based on the intervention received at their definitive fracture management surgery. Participants who do not receive one of the study interventions will be removed from this analysis. Similar to the primary analysis, we will use mixed effects regression models with a binomial distribution and the same covariates and correlation structure as the primary model. A more simplified structure will be considered if we encounter convergence issues with this model.

Missing Data: While we anticipate minimal missing outcome data, we will perform a sensitivity analysis on the primary and secondary analyses to explore the impact of missing outcome data. Our sensitivity analysis will be a complete case analysis, including only those patients with a known status of the outcome being analyzed.

Bayesian Analysis: The Bayesian analyses will be performed using four different priors (neutral with moderate strength, neutral flat, optimistic with moderate strength, and pessimistic with moderate strength) defined on a log-odds scale and described below. The neutral priors will be centered on a log odds of 0 (odds ratio of 1). The neutral flat prior will have a standard deviation of 100. The optimistic prior will be centered on the estimated effect size of a 0.64 odds ratio (log odds of -0.45). In contrast, the pessimistic prior is centered on the same effect size but for the alternative treatment. As suggested by Zampieri et al.,<sup>33</sup> the standard deviation of 0.44 was selected for the moderate strength priors as it allows for a 15% probability of the alternative treatment benefit in both the optimistic and pessimistic prior. The prior probability of our neutral prior with a moderate strength distribution implies a 68% chance the estimated effect will be between an odds

ratio of 0.64 and 1.36. The neutral prior with moderate strength will be our preferred prior in this sensitivity analysis.

286 Th287 a r288 tre

The modeling for the Bayesian analysis will be consistent with our primary analysis. We will use a mixed effects regression model with a Bernoulli distribution. The model will include time and treatment as fixed effects and use random effects to account for the complex correlation structure. The best fitting correlation structure will be determined using information criteria. If we experience convergence issues with this model structure, we will transition to a less complex model. We will report treatment effects as odds ratios with 95% credible intervals. We will also report the probability of treatment benefits of povidone-iodine, with 50% implying no difference in the probability of benefit between the two treatment groups.

## Priors used in the analysis with their interpretation and a visual depiction.

| Prior | Mean | Standard Deviation | Interpretation | Visualization |
|---|---|---|---|---|
| Neutral<br>with<br>moderate<br>strength | Log(1.00)<br>= 0 | 0.44 | "There is no strong information to suggest the intervention is good or bad in this study population, but we think extreme effect sizes are very unlikely." | Favors Povidone-Iodine Favors Chlorhexidine 0.8 0.4 0.0 0.22 0.82 1.38 0.83 0.83 0.83 0.83 0.84 0.85 |
| Neutral flat | Log(1.00)<br>= 0 | 100 | "None of the prior<br>research is relevant to<br>this trial, and we<br>cannot rule out<br>extreme effect sizes." | Favors Povidone-Iodine Favors Chlorhexidine 0.4 0.0 0.22 0.62 1 138 0.04 0.04 0.05 0.0 |

| Optimistic with moderate strength | Log(0.64)<br>= -0.45 | 0.44 | "We think povidone- iodine is more effective but cannot rule out that chlorhexidine is superior." | Favors Povidone-Iodine Favors Chlorhexidine 0.4 0.0 0.22 0.82 0.338 Odds Ratio |
|---|---|---|---|---|
| Pessimistic with moderate strength | Log(1.36) = 0.31 | 0.44 | "We think<br>chlorhexidine is more<br>effective but cannot<br>rule out that povidone-<br>iodine is superior." | Favors Povidone-Iodine Favors Chlorhexidine 1.2 Favors Povidone-Iodine Favors Chlorhexidine 0.8 0.8 0.8 0.8 0.8 0.8 0.8 0. |

297 **5.5 Harms** 

296

298

299

300

301

The number and percentage of patients experiencing serious adverse events will be presented by treatment arm. No formal statistical testing will be undertaken.

5.6 Statistical Software

The statistical analyses will be performed with SAS, version 9.4 (SAS Institute, Cary, NC) and R

(R Foundation for Statistical Computing, Vienna, Austria).

# 6.0 FIGURES AND TABLES

304

305

306 307

# **Table 1: Baseline characteristics**

| | Iodine Povacrylex in | Chlorhexidine in |
|---|---|---|
| | Alcohol | Alcohol |
| (3D) | (n= XX participants) | (n= XX participants) |
| Age, years, mean (SD) | | |
| Sex, n (%) | | |
| Female | | |
| Male | | |
| Prefer not to answer | | |
| Race or ethnicity, n (%) | | |
| White | | |
| Black | | |
| Central or South American | | |
| Asian | | |
| Indigenous | | |
| Native Hawaiian or Pacific Islander | | |
| Multiracial | | |
| Prefer not to answer | | |
| Body mass index, kg/m <sup>2</sup> , n (%) | | |
| Underweight (BMI < 18·5) | | |
| Normal weight $(18.5 - 24.9)$ | | |
| Overweight (25 – 29·9) | | |
| Obese (BMI > 30) | | |
| Diabetes, n (%) | | |
| Current smoker, n (%) | | |
| Injury severity score, mean (SD) | | |
| American Society of Anesthesiologist | | |
| Physical Score, n (%) | | |
| Class I or II | | |
| Class III or higher | | |
| Number of included closed fractures per | | |
| participant, n (%) | | |
| One | | |
| Two | | |
| Three | | |

309

310

311

312

313

314

315

**Table 2: Fracture Characteristics and Management** 

| Table 2: Fracture Characteristics and Man | Iodine Povacrylex in Alcohol (n= XX fractures) | Chlorhexidine in<br>Alcohol<br>(n= XX fractures) |
|---|---|---|
| Location of fracture, n (%) | | |
| Pelvis | | |
| Femur, proximal | | |
| Femur, shaft | | |
| Knee | | |
| Tibia, shaft | | |
| Tibia, distal | | |
| Foot and ankle | | |
| Periarticular fracture, n (%)* | | |
| Severe soft tissue injury, n (%)** | | |
| Temporary fracture stabilization, n (%) | | |
| Number of planned surgeries, n (%) | | |
| 1 | | |
| 2 | | |
| 3 | | |
| 4 | | |
| 5 or more | | |
| Duration of antibiotic administration (days), | | |
| median (IQR) | | |
| Closure method, n (%)*** | | |
| Primary wound closure | | |
| No closure attempted/secondary wound | | |
| healing | | |
| Skin graft | | |
| Local flap | | |
| Free flap | | |

<sup>\*</sup>Periarticular fractures are fractures of the distal femur, proximal tibia, distal tibia, or ankle.

<sup>\*\*</sup>Severe soft tissue injury is defined as having one of the following: 1) extensive skin contusion or crush injury, 2) severe damage to underlying muscle, 3) compartment syndrome, 4) degloving

<sup>\*\*\*</sup>More than one type of closure method may have been performed during surgery, but only the most complex method of closure is reported in the table using the following the hierarchy: 1) free flap, 2) local flap, 3) skin graft, 4) no closure attempted/secondary wound healing, 5) primary wound closure

316 **Table 3: Study outcomes** 

| | Iodine Povacrylex in<br>Alcohol (n=XXX)<br>number (%)* | Chlorhexidine in<br>Alcohol (n=XXX)<br>number (%)* | Odds<br>Ratio**<br>(95% CI) | p-value** | Risk<br>Difference**<br>(95% CI) |
|---|---|---|---|---|---|
| Primary outcome | n=XXX | n=XXX | (9376 CI) | | (93% CI) |
| Surgical site infection | | | | | |
| Superficial infection | | | | | |
| Deep incisional | | | | | |
| Organ/space infection | | | | | |
| | | | • | | |
| Alternative definitions of surgical site | n=XXX | n=XXX | | | |
| infection | | | | | |
| Any surgical site infection by 365 | | | | | |
| days | | | | | |
| Fracture-related infection by 365 days | | | | | |
| Secondary outcome | n=XXX | n=XXX | | | |
| Unplanned reoperation by 365 days | | | | | |
| Unplanned reoperation for infection | | | | | |
| by 365 days | | | | | |
| Unplanned reoperation for wound | | | | | |
| healing complications by 365 days | | | | | |
| Unplanned reoperation to promote | | | | | |
| fracture healing by 365 days | | | | | |

CI = Confidence Interval

<sup>317</sup> 318 319 \*Percentages based on complete case description

\*\*Missing outcome data were imputed using multiple imputations



## 1 Figure 2. Forest plot of subgroup analyses



## LIST OF ABBREVIATIONS

4 5

3

ASC/AST Active surveillance culture/testing

PREPARE A Pragmatic Randomized trial Evaluating Pre-operative Alcohol

skin solutions in FRactured Extremities

BMI Body mass index

CDC Centers for Disease Control

FRI Fracture-related infection

ST Soft tissue

SSI Surgical site infection

6

7

8

9 **DECLARATIONS** 10 **Ethics Approval and Consent to Participate** 11 12 Ethics approval has been obtained from the Hamilton Integrated Research Ethics Board for the 13 Methods Center (#4336), the Advarra Central Institutional Review Board (formerly Chesapeake 14 Institutional Review Board) (#Pro00023709), and each clinical site's local institutional review 15 board or research ethics board, if they are not using the central institutional review board. Written 16 informed consent has been obtained for study participation. 17 18 **Consent for Publication** 19 Not applicable 20 21 **Availability of Data and Materials** 22 The datasets generated and/or analyzed during the current study are not publicly available due to 23 the trial still being ongoing, but will be available from the corresponding author on reasonable 24 request. 25 26 **Competing Interests** 27 Dr. Slobogean reports editorial or governing board for the Journal of Orthopaedic Trauma, board 28 or committee member for the Orthopaedic Trauma Association, paid consultant for Smith & 29 Nephew, and paid consultant for Zimmer, all outside the submitted work. Dr. Sprague reports 30 board or committee member for Orthopaedic Trauma Association, employment from Global 31 Research Solutions Inc. and consultant fees from the University of Sherbrooke and Platform Life 32 Sciences, all outside the submitted work. Dr. Bhandari reports paid consultant from AgNovos

- Healthcare, research support from the Canadian Institutes of Health Research (CIHR), board or committee member for the International Society of Orthopaedic Surgery and Traumatology (SICOT), research support from the National Institutes of Health (NIAMS & NICHD), research support from Physicians' Services Incorporated, paid consultant for Sanofi-Aventis, paid consultant for Smith & Nephew, and research support from the U.S. Department of Defense, all outside the submitted work. Dr. O'Hara reports stock or stock options from Arbutus Medical Inc,
- 41 Funding

40

44

48

51

56

- The PREPARE trial is funded by the Patient-Centered Outcomes Research Institute (PCS-1609-
- 43 36512) and the Canadian Institutes of Health Research (Foundation Grant).

all outside the submitted work. All other authors have nothing to report.

- 45 Authors' Contributions
- 46 All authors have been major contributors in writing the statistical analysis plan. All authors have
- 47 read and approved the statistical analysis plan.
- 49 Acknowledgements
- 50 **PREP-IT Investigators**
- 52 Executive Committee: Gerard P. Slobogean (Principal Investigator, University of Maryland
- 53 School of Medicine, Baltimore, MD); Sheila Sprague (Principal Investigator, McMaster
- 54 University, Hamilton, ON); Jeffrey L. Wells (Patient Representative, Trauma Survivors Network,
- Falls Church, VA); Mohit Bhandari (Principal Investigator, McMaster University, Hamilton, ON)
- 57 Steering Committee: Gerard P. Slobogean (Co-Chair, University of Maryland School of
- Medicine, Baltimore, MD); Mohit Bhandari (Co-Chair, McMaster University, Hamilton, ON);
- 59 Sheila Sprague (Principal Investigator, McMaster University, Hamilton, ON); Anthony D. Harris
- 60 (University of Maryland School of Medicine, Baltimore, MD); C. Daniel Mullins (University of
- Maryland School of Medicine, Baltimore, MD); Lehana Thabane (McMaster University,

Hamilton, ON); Jeffrey L. Wells (Trauma Survivors Network, Falls Church, VA); Amber Wood (Association of periOperative Registered Nurses, Denver, CO)

Adjudication Committee: Gregory J. Della Rocca (Chair, University of Missouri, Columbia, MO); Anthony D. Harris (University of Maryland School of Medicine, Baltimore, MD); Joan N. Hebden (University of Maryland School of Medicine, Baltimore, MD); Kyle J. Jeray (Prisma Health - Upstate, Greenville, SC); Lucas S. Marchand (University of Utah, Salt Lake City, UT); Lyndsay M. O'Hara (University of Maryland School of Medicine, Baltimore, MD); Robert D. Zura (LSU Health, New Orleans, LA); Christopher Lee (University of California, Los Angeles, CA); Joseph T. Patterson (University of Southern California, Los Angeles, CA)

**Data and Safety Monitoring Committee:** Michael J. Gardner (Chair, Stanford University School of Medicine, Palo Alto, CA); Jenna Blasman (Patient Representative, Kitchener, ON); Jonah Davies (University of Washington, Seattle, WA); Stephen Liang (Washington University, St. Louis, MO); Monica Taljaard (Ottawa Hospital Research Institute, Ottawa, ON)

**Research Methodology Core:** PJ Devereaux (McMaster University, Hamilton, ON); Gordon Guyatt (McMaster University, Hamilton, ON); Lehana Thabane (McMaster University, Hamilton, ON); Diane Heels-Ansdell (McMaster University, Hamilton, ON)

Patient Centred Outcomes Core: Debra Marvel (Patient Representative, Baltimore, MD); Jana E. Palmer (Patient Representative, Baltimore, MD); Jeffrey L. Wells (Patient Representative, Trauma Survivors Network, Falls Church, VA); Jeff Friedrich (Editor, Slate Magazine, Washington, DC); C. Daniel Mullins (University of Maryland School of Medicine, Baltimore, MD); Nathan N. O'Hara (University of Maryland School of Medicine, Baltimore, MD); Frances Grissom (Trauma Survivor Network, Baltimore, MD)

**Orthopaedic Surgery Core:** Gregory J. Della Rocca (University of Missouri, Columbia, MO); I. Leah Gitajn (Dartmouth University, Hanover, NH); Kyle J. Jeray (Prisma Health - Upstate, Greenville, SC); Saam Morshed (San Francisco General Hospital, San Francisco, CA); Robert V. O'Toole (University of Maryland School of Medicine, Baltimore, MD); Bradley Petrisor (Hamilton Health Sciences, Hamilton, ON)

Operating Room Core: Franca Mossuto (Hamilton Health Sciences, Hamilton, ON)
Infectious Disease Core: Anthony D. Harris (University of Maryland School of Medicine, Baltimore, MD); Manjari G. Joshi (University of Maryland School of Medicine, Baltimore, MD)

**Military Core:** Jean-Claude G. D'Alleyrand (Walter Reed National Military Medical Center, 100 Bethesda, MD); Justin Fowler (United States Army, USA); Jessica C. Rivera (San Antonio 101 Military Medical Center, San Antonio, TX); Max Talbot (Canadian Armed Forces, Montreal, QC)

- McMaster University Methods Center (Hamilton, ON): Sheila Sprague (Principal Investigator);
   Mohit Bhandari (Principal Investigator); David Pogorzelski (Research Coordinator); Shannon
- Dodds (Research Coordinator); Silvia Li (Research Coordinator); Gina Del Fabbro (Research
- 106 Assistant); Olivia Paige Szasz (Research Assistant); Diane Heels-Ansdell (Statistician); Paula

- 107 McKay (Manager); Alexandra Minea (Research Coordinator); Kevin Murphy (Research
- 108 Assistant); Sofia Bzovsky (Statistical Analyst)
- 110 University of Maryland School of Medicine Administrative Center (Baltimore, MD): Gerard
- P. Slobogean (Principal Investigator); Nathan N. O'Hara (Manager); Andrea L. Howe (Project
- Manager); Haley Demyanovich (Project Manager), Wayne Hoskins (Co-Investigator)
- 114 University of Maryland School of Pharmacy, The PATIENTS Program (Baltimore, MD): C.
- Daniel Mullins (Executive Director); Michelle Medeiros (Director of Research); Genevieve Polk
- 116 (Assistant Director, Dissemination and Research); Eric Kettering (Senior Instructional Technology
- and Dissemination Specialist); Nirmen Mahal (Program Specialist)
- 119 **PREP-IT Clinical Sites:**

113

118

126

131

143

148

151

- 120 Lead Clinical Site (Aqueous-PREP and PREPARE):
- 121 University of Maryland School of Medicine, R Adams Cowley Shock Trauma Center,
- Baltimore, MD: Robert V. O'Toole, Jean-Claude G. D'Alleyrand, Andrew Eglseder, Aaron
- 123 Johnson, Christopher Langhammer, Christopher Lebrun, Jason Nascone, Raymond Pensy,
- 124 Andrew Pollak, Marcus Sciadini, Gerard P. Slobogean, Yasmin Degani, Haley K. Demyanovich,
- 125 Andrea L. Howe, Nathan N. O'Hara, Heather Phipps, Eric Hempen
- 127 Aqueous-PREP and PREPARE:
- Hamilton Health Sciences General Site, Hamilton, ON: Bradley Petrisor, Herman Johal, Bill
- Ristevski, Dale Williams, Matthew Denkers, Krishan Rajaratnam, Jamal Al-Asiri, Jodi L. Gallant,
- 130 Kaitlyn Pusztai, Sarah MacRae, Sara Renaud.
- 132 **Prisma Health Upstate, Greenville, SC**: Kyle J. Jeray, John D. Adams, Michael L. Beckish,
- 133 Christopher C. Bray, Timothy R. Brown, Andrew W. Cross, Timothy Dew, Gregory K. Faucher,
- Richard W. Gurich Jr, David E. Lazarus, S. John Millon, M. Christian Moody, M. Jason Palmer,
- Scott E. Porter, Thomas M. Schaller, Michael S. Sridhar, John L. Sanders, L. Edwin Rudisill, Jr.
- Michael J. Garitty, Andrew S. Poole, Michael L. Sims, Clark M. Walker, Robert Carlisle, Erin A.
- Hofer, Brandon Huggins, Michael Hunter, William Marshall, Shea B. Ray, Cory Smith, Kyle M.
- Altman, Erin Pichiotino, Julia C. Quirion, Markus F. Loeffler, Erin R. Pichiotino, Austin A. Cole,
- Ethan J. Maltz, Wesley Parker, T. Bennett Ramsey, Alex Burnikel, Michael Colello, Russell
- 140 Stewart, Jeremy Wise, Matthew Anderson, Joshua Eskew, Benjamin Judkins, James M. Miller,
- 141 Stephanie L. Tanner, Rebecca G. Snider, Christine E. Townsend, Kayla H. Pham, Abigail Martin,
- Emily Robertson, Emily Bray, J. Wilson Sykes, Krystina Yoder, Kelsey Conner, Harper Abbott
- 144 IU Health Methodist Hospital, Indianapolis, IN: Roman M. Natoli, Todd O. McKinley, Walter
- W. Virkus, Anthony T. Sorkin, Jan P. Szatkowski, Brian H. Mullis, Yohan Jang, Luke A. Lopas,
- Lauren C. Hill, Courteney L. Fentz, Maricela M. Diaz, Krista Brown, Katelyn M. Garst, Emma
- 147 W. Denari
- 149 San Antonio Military Medical Center, San Antonio, TX: Patrick Osborn, Justin Fowler, Sarah
- N. Pierrie, Bradley Kessler, Maria Herrera

- 152 University of California, San Francisco, San Francisco, CA: Saam Morshed, Theodore
- 153 Miclau, Meir T. Marmor, Amir Matityahu, R. Trigg McClellan, David Shearer, Paul Toogood,
- Anthony Ding, Jothi Murali, Ashraf El Naga, Jennifer Tangtiphaiboontana, Tigist Belaye, Eleni
- 155 Berhaneselase, Dmitry Pokhvashchev
- 156
- 157 Aqueous-PREP:
- Vanderbilt Medical Center, Nashville, TN: William T. Obremskey, Amir Alex Jahangir, Manish
- 159 Sethi, Robert Boyce, Daniel J. Stinner, Phillip P. Mitchell, Karen Trochez, Elsa Rodriguez, Charles
- 160 Pritchett, Natalie Hogan, A. Fidel Moreno

- 162 University of Florida, Gainesville, FL: Jennifer E. Hagen, Matthew Patrick, Richard Vlasak,
- 163 Thomas Krupko, Michael Talerico, Marybeth Horodyski, Marissa Pazik, Elizabeth Lossada-Soto

164

- 165 McGovern Medical School at UTHealth Houston, Houston, TX: Joshua L. Gary, Stephen J.
- Warner, John W. Munz, Andrew M. Choo, Timothy S. Achor, Milton L. "Chip" Routt, Michael
- 167 Kutzler, Sterling Boutte, Ryan J. Warth

168

- Wright State University, Dayton, OH: Michael J. Prayson, Indresh Venkatarayappa, Brandon
- Horne, Jennifer Jerele, Linda Clark

171

- 172 Banner University Medical Center Tucson, Tucson, AZ: Christina Boulton, Jason Lowe,
- John T. Ruth, Brad Askam, Andrea Seach, Alejandro Cruz, Breanna Featherston, Robin Carlson,
- 174 Iliana Romero, Isaac Zarif

175

- 176 The CORE Institute, Phoenix, AZ: Niloofar Dehghan, Michael McKee, Clifford B. Jones, Debra
- 177 L. Sietsema, Alyse Williams, Tayler Dykes

178

- 179 Vall d'Hebron University Hospital, Barcelona, Spain: Ernesto Guerra-Farfan, Jordi Tomas-
- Hernandez, Jordi Teixidor-Serra, Vicente Molero-Garcia, Jordi Selga-Marsa, Juan Antonio
- Porcel-Vazquez, Jose Vicente Andres-Peiro, Ignacio Esteban-Feliu, Nuria Vidal-Tarrason, Jordi
- 182 Serracanta, Jorge Nuñez-Camarena, Maria del Mar Villar-Casares, Jaume Mestre-Torres, Pilar
- 183 Lalueza-Broto, Felipe Moreira-Borim, Yaiza Garcia-Sanchez

184

- 185 Hospital Universitari Parc Tauli, Barcelona, Spain: Francesc Marcano-Fernández, Laia
- Martínez-Carreres, David Martí-Garín, Jorge Serrano-Sanz, Joel Sánchez-Fernández, Matsuyama
- 187 Sanz-Molero, Alejandro Carballo, Xavier Pelfort, Francesc Acerboni-Flores, Anna Alavedra-
- 188 Massana, Neus Anglada-Torres, Alexandre Berenguer, Jaume Cámara-Cabrera, Ariadna
- Caparros-García, Ferran Fillat-Gomà, Ruben Fuentes-López, Ramona Garcia-Rodriguez, Nuria
- 190 Gimeno-Calavia, Marta Martínez-Álvarez, Patricia Martínez-Grau, Raúl Pellejero-García, Ona
- 191 Ràfols-Perramon, Juan Manuel Peñalver, Mònica Salomó Domènech, Albert Soler-Cano, Aldo
- 192 Velasco-Barrera, Christian Yela-Verdú, Mercedes Bueno-Ruiz, Estrella Sánchez-Palomino, Vito
- 193 Andriola, Matilde Molina-Corbacho, Yeray Maldonado-Sotoca, Alfons Gasset-Teixidor, Jorge
- 194 Blasco-Moreu, Núria Fernández-Poch, Josep Rodoreda-Puigdemasa, Arnau Verdaguer-Figuerola,
- 195 Heber Enrique Cueva-Sevieri, Santiago Garcia-Gimenez

196

197 PREPARE:

- 198 FRASER HEALTH AUTHORITY/Royal Columbian Hospital, New Westminster, BC:
- Darius G. Viskontas, Kelly L. Apostle, Dory S. Boyer, Farhad O. Moola, Bertrand H. Perey,
- Trevor B. Stone, H. Michael Lemke, Ella Spicer, Kyrsten Payne
- 201
- 202 Inova Fairfax Medical Campus, Falls Church, VA: Robert A. Hymes, Cary C. Schwartzbach,
- Jeff E. Schulman, A. Stephen Malekzadeh, Michael A. Holzman, Greg E. Gaski, Jonathan Wills,
- 204
- Wake Forest Baptist Health, Winston-Salem, NC: Holly Pilson, Eben A. Carroll, Jason J.
- Halvorson, Sharon Babcock, J. Brett Goodman, Martha B. Holden, Wendy Williams, Taylor Hill,
- 207 Ariel Brotherton
- 208
- 209 MetroHealth Medical Center, Cleveland, OH: Nicholas M. Romeo, Heather A. Vallier, Anna
- 210 Vergon
- 211
- 212 University of Utah, Salt Lake City, Utah: Thomas F. Higgins, Justin M. Haller, David L.
- 213 Rothberg, Lucas S. Marchand, Zachary M. Olsen, Abby V. McGowan, Sophia Hill, Morgan K.
- 214 Dauk
- 215
- 216 University of Mississippi Medical Center, Jackson, MS: Patrick F. Bergin, George V. Russell,
- 217 Matthew L. Graves, John Morellato, Sheketha L. McGee, Eldrin L. Bhanat, Ugur Yener, Rajinder
- 218 Khanna, Priyanka Nehete
- 219
- 220 Sanford Health, Sioux Falls, SD: David Potter, Robert VanDemark III, Kyle Seabold, Nicholas
- 221 Staudenmier
- 222
- 223 Dartmouth-Hitchcock Medical Center, Lebanon, NH: I. Leah Gitajn, Marcus Coe, Kevin
- Dwyer, Devin S. Mullin, Theresa A. Chockbengboun, Peter A. DePalo Sr.
- 225
- 226 Carolinas Medical Center, Atrium Health Musculoskeletal Institute, Charlotte, NC: Kevin
- 227 Phelps, Michael Bosse, Madhay Karunakar, Laurence Kempton, Stephen Sims, Joseph Hsu,
- 228 Rachel Seymour, Christine Churchill, Ada Mayfield, Juliette Sweeney
- 229
- 230 University of Maryland, Capital Region Health: Largo, MD: Todd Jaeblon, Robert Beer, Haley
- K. Demyanovich, Brent Bauer, Sean Meredith, Sneh Talwar
- 232
- 233 University of Wisconsin Madison, Madison, WI: Christopher M. Domes
- 234
- Duke University Hospital, Durham, NC: Mark J. Gage, Rachel M. Reilly, Ariana Paniagua,
- JaNell Dupree
- 237
- 238 Brigham Women's Hospital, Boston, MA: Michael J. Weaver, Arvind G. von Keudell, Abigail
- E. Sagona
- 240
- 241 University of Pennsylvania, Philadelphia, PA: Samir Mehta, Derek Donegan, Annamarie
- 242 Horan, Mary Dooley
- 243

| 244 | Massachusetts General Hospital, Boston, MA: Marilyn Heng, Mitchel B. Harris, David W. |
|---|---|
| 245 | Lhowe, John G. Esposito, Ahmad Alnasser |
| 246 | |
| 247 | Bryan Medical Center, Lincoln, Nebraska: Steven F. Shannon, Alesha N. Scott, Bobbi Clinch, |
| 248 | Becky Weber |
| 249 | |
| 250 | University of Cincinnati, Cincinnati, OH: Michael J. Beltran, Michael T. Archdeacon, Henry |
| 251 | Claude Sagi, John D. Wyrick, Theodore Toan Le, Richard T. Laughlin, Cameron G. Thomson, |
| 252 | Kimberly Hasselfeld |
| 253 | |
| 254 | Cedars-Sinai Medical Center, Los Angeles, CA: Carol A. Lin, Mark S. Vrahas, Charles N. |
| 255 | Moon, Milton T. Little, Geoffrey S. Marecek, Denice M. Dubuclet |
| 256 | |
| 257 | University of California, Irvine, Orange, CA: John A. Scolaro, James R. Learned, Philip K. |
| 258 | Lim, Susan Demas, Arya Amirhekmat, Yan Marco Dela Cruz |
| 259 | |
| 260 | |
| 261 | |

REFERENCES

262

- Centers for Disease Control and Prevention (CDC). Surgical Site Infection (SSI) Event.;
   2017.
- 265 2. Darouiche RO, Wall MJ, Itani KMF, et al. Chlorhexidine-Alcohol versus Povidone-Iodine for Surgical-Site Antisepsis. *N Engl J Med*. 2010;362(1):18-26.
- Tuuli MG, Liu J, Stout MJ, et al. A Randomized Trial Comparing Skin Antiseptic Agents at Cesarean Delivery. *N Engl J Med*. 2016;374(7):647-655.
- Swenson BR, Sawyer RG. Importance of alcohol in skin preparation protocols. *Infect Control Hosp Epidemiol*. 2010;31(9):977.
- 5. Swenson BR, Hedrick TL, Metzger R, Bonatti H, Pruett TL, Sawyer RG. Effects of preoperative skin preparation on postoperative wound infection rates: a prospective study of 3 skin preparation protocols. *Infect Control Hosp Epidemiol*. 2009;30(10):964-971.
- FLOW Investigators, Bhandari M, Jeray KJ, et al. A Trial of Wound Irrigation in the Initial
   Management of Open Fracture Wounds. N Engl J Med. 2015;373(27):2629-2641.
   doi:10.1056/NEJMoa1508502
- 7. Gamble C, Krishan A, Stocken D, et al. Guidelines for the Content of Statistical Analysis Plans in Clinical Trials. *JAMA*. 2017;318(23):2337. doi:10.1001/jama.2017.18556
- Dwan K, Li T, Altman DG, Elbourne D. CONSORT 2010 statement: extension to randomised crossover trials. *BMJ*. Published online July 31, 2019:l4378.
   doi:10.1136/bmj.l4378
- 9. Sprague S, Scott T, Dodds S, et al. Cluster identification, selection, and description in cluster randomized crossover trials: the PREP-IT trials. *Trials*. 2020;21(1):712.
- 10. Fergusson D, Aaron SD, Guyatt G, Hébert P. Post-randomisation exclusions: the intention to treat principle and excluding patients from analysis. *BMJ*. 2002;325(7365):652-654. doi:10.1136/bmj.325.7365.652
- Ibrahim DA, Swenson A, Sassoon A, Fernando ND. Classifications In Brief: The Tscherne
   Classification of Soft Tissue Injury. *Clin Orthop*. 2017;475(2):560-564.
   doi:10.1007/s11999-016-4980-3
- 290 12. FLOW Investigators, Bhandari M, Jeray KJ, et al. A Trial of Wound Irrigation in the Initial Management of Open Fracture Wounds. *N Engl J Med*. 2015;373(27):2629-2641.
- 292 13. FAITH Investigators. Fracture fixation in the operative management of hip fractures (FAITH): an international, multicentre, randomised controlled trial. *Lancet Lond Engl.* 2017;389(10078):1519-1527. doi:10.1016/S0140-6736(17)30066-1
- 295 14. HEALTH Investigators, Bhandari M, Einhorn TA, et al. Total Hip Arthroplasty or
- Hemiarthroplasty for Hip Fracture. N Engl J Med. 2019;381(23):2199-2208.
- 297 doi:10.1056/NEJMoa1906190
- 298 15. the CONSORT Group, Schulz KF, Altman DG, Moher D. CONSORT 2010 Statement:
- updated guidelines for reporting parallel group randomised trials. *Trials*. 2010;11(1):32.
- 300 doi:10.1186/1745-6215-11-32
- 301 16. Morgan KE, Forbes AB, Keogh RH, Jairath V, Kahan BC. Choosing appropriate analysis
- methods for cluster randomised cross-over trials with a binary outcome: K. E. MORGAN
- 303 ET AL. Stat Med. 2017;36(2):318-333. doi:10.1002/sim.7137
- 304 17. Hemming K, Kasza J, Hooper R, Forbes A, Taljaard M. A tutorial on sample size
- calculation for multiple-period cluster randomized parallel, cross-over and stepped-wedge
- trials using the Shiny CRT Calculator. *Int J Epidemiol*. 2020;49(3):979-995.
- 307 doi:10.1093/ije/dyz237
- 308 18. Hemming K, Taljaard M, Weijer C, Forbes AB. Use of multiple period, cluster randomised,
- crossover trial designs for comparative effectiveness research. *BMJ*. Published online
- November 4, 2020:m3800. doi:10.1136/bmj.m3800
- 311 19. Wise BT, Connelly D, Rocca M, et al. A Predictive Score for Determining Risk of Surgical
- 312 Site Infection After Orthopaedic Trauma Surgery. *J Orthop Trauma*. 2019;33(10):506-513.
- 313 doi:10.1097/BOT.000000000001513
- 314 20. Thompson DD, Lingsma HF, Whiteley WN, Murray GD, Steyerberg EW. Covariate
- adjustment had similar benefits in small and large randomized controlled trials. *J Clin*
- 316 Epidemiol. 2015;68(9):1068-1075. doi:10.1016/j.jclinepi.2014.11.001
- 21. Program of Randomized Trials to Evaluate Pre-operative Antiseptic Skin Solutions in
- Orthopaedic Trauma (PREP-IT) Investigators, Slobogean GP, Sprague S, et al.
- 319 Effectiveness of Iodophor vs Chlorhexidine Solutions for Surgical Site Infections and
- 320 Unplanned Reoperations for Patients Who Underwent Fracture Repair: The PREP-IT
- 321 Master Protocol. *JAMA Netw Open.* 2020;3(4):e202215.
- 322 22. Campbell MK, Piaggio G, Elbourne DR, Altman DG, CONSORT Group. Consort 2010
- statement: extension to cluster randomised trials. *BMJ*. 2012;345:e5661.
- 324 doi:10.1136/bmj.e5661
- 325 23. Rubin DB. Multiple imputation for survey nonresponse. Published online 1987.
- 326 24. Wang R, Lagakos SW, Ware JH, Hunter DJ, Drazen JM. Statistics in medicine--reporting
- of subgroup analyses in clinical trials. *N Engl J Med*. 2007;357(21):2189-2194.
- 328 25. Sun X, Ioannidis JPA, Agoritsas T, Alba AC, Guyatt G. How to use a subgroup analysis:
- users' guide to the medical literature. JAMA. 2014;311(4):405-411.

- 330 26. Sun X, Briel M, Walter SD, Guyatt GH. Is a subgroup effect believable? Updating criteria to evaluate the credibility of subgroup analyses. *BMJ*. 2010;340:c117.
- 332 27. Sun X, Briel M, Busse JW, et al. Subgroup Analysis of Trials Is Rarely Easy (SATIRE): a
- study protocol for a systematic review to characterize the analysis, reporting, and claim of subgroup effects in randomized trials. *Trials*. 2009;10:101.
- 335 28. Schandelmaier S, Briel M, Varadhan R, et al. Development of the Instrument to assess the
- Credibility of Effect Modification Analyses (ICEMAN) in randomized controlled trials and
- meta-analyses. CMAJ Can Med Assoc J J Assoc Medicale Can. 2020;192(32):E901-E906.
- 338 doi:10.1503/cmaj.200077
- 339 29. Metsemakers Wj, Morgenstern M, McNally MA, et al. Fracture-related infection: A
- consensus on definition from an international expert group. *Injury*. 2018;49(3):505-510.
- 341 doi:10.1016/j.injury.2017.08.040
- 342 30. Metsemakers WJ, Morgenstern M, McNally MA, et al. Fracture-related infection: A
- consensus on definition from an international expert group. *Injury*. 2018;49:505-510.
- 34. Metsemakers WJ, Kuehl R, Moriarty TF, et al. Infection after fracture fixation: Current
- surgical and microbiological concepts. *Injury*. 2018;49(3):511-522.
- 346 32. Study to Prospectively Evaluate Reamed Intramedullary Nails in Patients with Tibial
- Fractures Investigators, Bhandari M, Guyatt G, et al. Randomized Trial of Reamed and
- 348 Unreamed Intramedulary Nailing of Tibial Shaft Fractures. *J Bone Jt Surg-Am Vol.*
- 349 2008;90(12):2567-2578.
- 350 33. Zampieri FG, Casey JD, Shankar-Hari M, Harrell FE, Harhay MO. Using Bayesian
- Methods to Augment the Interpretation of Critical Care Trials. An Overview of Theory and
- Example Reanalysis of the Alveolar Recruitment for Acute Respiratory Distress Syndrome
- 353 Trial. Am J Respir Crit Care Med. 2021;203(5):543-552. doi:10.1164/rccm.202006-
- 354 2381CP

# A <u>Pragmatic Randomized trial Evaluating Pre-operative</u> <u>Alcohol skin solutions in <u>FRactured Extremities</u> (PREPARE Open): Statistical Analysis Plan</u>

**Trial Registration:** clinicaltrials.gov, NCT03523962. Registered May 14, 2018, https://clinicaltrials.gov/ct2/show/NCT03523962

**SAP Version:** 1.0

**Protocol Version: 2.2** 

**SAP Revisions:** None

**Disclaimer:** This SAP was adapted from the Aqueous-PREP (Aqueous skin antisepsis before surgical fixation of open fractures) SAP, which was published in *Trials* in September 2022 (https://trialsjournal.biomedcentral.com/articles/10.1186/s13063-022-06541-0). A copy of the Aqueous-PREP SAP was also uploaded onto the ClinicalTrials.gov trial registration page (https://clinicaltrials.gov/ct2/show/NCT03385304). The Aqueous-PREP primary manuscript was published in *The Lancet* in October 2022 (https://www.thelancet.com/journals/lancet/article/PIIS0140-6736(22)01652-X/fulltext#seccestitle200).

| Reviewed and Approved by: | | |
|---|---|---|
| Dr. Gerard Slobogean<br>(Principal Investigator) | Signature: Occusioned by: 61 crard Slobogean 7DFE42965445427 | Date: 22-Feb-2023 |
| Dr. Sheila Sprague<br>(Principal Investigator) | Signature: | Date: 21-Feb-2023 |
| Dr. Nathan N. O'Hara<br>(Statistician) | Signature: Nathan O'Hara | Date: 21-Feb-2023 |
| Diane Heels-Ansdell<br>(Statistician) | Signature: Docusigned by: | Date: 27-Feb-2023 |
| Sofia Bzovsky<br>(Statistical Analyst) | Signature: Sofia Bousky | Date: 21-Feb-2023 |

#### **ABSTRACT**

## **Background**

Approximately 1 in 10 patients with a surgically treated open fracture will develop a surgical site infection. The PREPARE Open trial will investigate the effect of iodine povacrylex (0.7% free iodine) in 74% isopropyl alcohol versus 2% chlorhexidine gluconate in 70% isopropyl alcohol antiseptic solutions in reducing infections after open fracture surgery. The study protocol was published in April 2020.

#### **Methods and Design**

The PREPARE Open trial is a pragmatic, multicentre, open-label, randomized multiple period cluster crossover trial. Each participating cluster is randomly assigned in a 1:1 ratio to provide 1 of the 2 study interventions on all eligible patients during a study period. The intervention periods are 2 months in length. After completing a 2-month period, the participating cluster crosses over to the alternative intervention. We plan to enroll a minimum of 1540 patients at 22 sites.

## Results

The primary outcome is surgical site infection guided by the Centers for Disease Control and Prevention's National Healthcare Safety Network reporting criteria (2017). All participants' surgical site infection surveillance period will end 30 days after definitive fracture management surgery for superficial infections and 90 days after definitive fracture management surgery for deep incisional or organ/space infections. The secondary outcome is an unplanned fracture-related reoperation within 12 months of the fracture.

## Conclusion

This manuscript serves as the formal statistical analysis plan (version 1.0) for the PREPARE Open trial. The statistical analysis plan was completed on February 21, 2023.

# Keywords

Open fracture, surgical site infection, alcohol antiseptic solutions

#### 1.0 INTRODUCTION

## 1.1 Background and Rationale

The prevention of infection is a critical goal of perioperative care for patients with surgically treated open fractures. Surgical site infections are often devastating complications for open fracture patients because of the unplanned reoperations, fracture healing difficulties, and adverse events from prolonged antibiotic treatments. Given the severity of open fractures, maximizing the effectiveness of current prophylactic procedures is essential.

Standard practice in the management of open fractures includes cleaning the injured limb with an antiseptic skin solution in the operating room prior to making a surgical incision. The available solutions kill bacteria and decrease the quantity of native skin flora, thereby reducing surgical site infection.<sup>2–5</sup> While there is extensive guidance on specific procedures for prophylactic antibiotic use and standards for sterile technique, the evidence regarding the choice of antiseptic skin preparation solution is very limited for open fracture surgery.

The PREPARE Open trial will provide the necessary evidence to guide the choice of antiseptic skin solution to prevent surgical site infections in patients with open fractures. The trial is poised to significantly impact the care and outcomes of open extremity fracture patients.

## 1.2 Objectives

The overall objective of the PREPARE Open trial is to compare the effect of iodine povacrylex (0.7% free iodine) in 74% isopropyl alcohol versus 2% chlorhexidine gluconate in 70% isopropyl alcohol antiseptic solutions for the surgical management of open fractures.

Primary Objective and Hypothesis

To determine the effect of iodine povacrylex (0.7% free iodine) in 74% isopropyl alcohol versus 2% chlorhexidine gluconate in 70% isopropyl alcohol antiseptic solutions in preventing surgical site infections. We hypothesize that iodine povacrylex in alcohol antiseptic will be more effective in preventing surgical site infections than chlorhexidine gluconate in alcohol antiseptic.<sup>5,6</sup>

Secondary Objective and Hypothesis

To determine the effect of iodine povacrylex (0.7% free iodine) in 74% isopropyl alcohol versus 2% chlorhexidine gluconate in 70% isopropyl alcohol antiseptic solutions in preventing unplanned fracture-related reoperations. We hypothesize that iodine povacrylex in alcohol antiseptic will be more effective in preventing unplanned reoperations than chlorhexidine gluconate in alcohol antiseptic.<sup>5,6</sup>

Subgroup Objectives and Hypotheses

We will perform three subgroup analyses to determine if the effects of preoperative antiseptic skin solutions on surgical site infection vary within clinically relevant subgroups. The subgroups will be defined by i) the severity of the open fracture; ii) the location of the fracture; and iii) the severity of wound contamination. We hypothesize that the magnitude of the effect of iodine povacrylex (0.7% free iodine) in 74% isopropyl alcohol compared with 2% chlorhexidine gluconate in 70% isopropyl alcohol antiseptic in preventing surgical site infections will be greater in Gustilo-Anderson type III open fractures versus Gustilo-Anderson type I or II open fractures, lower extremity fractures versus upper extremity fractures, and wounds with embedded contamination

versus wounds with no, minimal, or surface contamination according to the Orthopaedic Trauma Association Open Fracture Classification (OTA-OFC).<sup>8–10</sup>

## 1.3 Reporting

The structure of this statistical analysis plan follows the Guidelines for the Content of Statistical Analysis Plans in Clinical Trials.<sup>11</sup> The reporting of the trial results will follow the 2010 CONSORT statement and the extension statements for Cluster Trials and Randomized Crossover Trials, as applicable.<sup>12</sup> Additional statistical analyses plans will be developed for secondary analyses of the trial data.

#### 2.0 STUDY METHODS

## 2.1 Trial Design

1

2

9

10

17

18

- 3 The study is a pragmatic, multicentre, open-label, randomized multiple period cluster crossover
- 4 trial. We defined clusters as orthopaedic practices within participating hospitals, with each
- 5 participating hospital having only one participating orthopaedic practice. 13 The intervention
- 6 periods are approximately 2 months in length. After completing a 2-month period, the participating
- 7 cluster crosses over to the alternative intervention where they use the other study solution for the
- 8 next 2-month period. There are no washout periods between treatment periods.

## 2.2 Randomization

- 11 The order of treatment allocation for each orthopaedic practice (cluster) will be randomly assigned
- using a computer-generated randomization table. Each cluster will start with the initially allocated
- study solution and crossover to the other solution for their second recruitment period. This process
- of alternating treatments will repeat approximately every 2 months as dictated by the initial
- 15 randomization until enrollment targets are met. The randomization will be in a 1:1 ratio,
- unrestricted, and executed only prior to the first sequence.

## 2.3 Sample Size

- 19 A sample size of 1540 patients will have 80% power to detect a 38% reduction in the odds of
- 20 infection with a two-sided alpha of 0.05. This estimate allows for a 10% loss to follow-up and
- assumes a baseline infection risk of 12.5%, 10 recruiting clusters, no between-period variance, and
- a 0.095 between-cluster variance. After the initial power calculations, we determined that
- 23 additional clusters were required to meet the study timelines. As such, we increased the number of

24 clusters from 10 to a minimum of 22. The increase in clusters results in a marginal increase in 25 statistical power (approximately 2%). 26 27 2.4 Framework 28 All study outcomes will be tested for superiority. 29 30 2.5 Interim Analysis and Stopping Guidance 31 PREPARE Open does not have a planned interim analysis. However, the trial's Data and Safety 32 Monitoring Committee reviews the reporting of serious adverse events biannually and can 33 recommend early stopping if safety concerns are identified. 34 35 2.6 Timing of Outcome Assessments 36 Research personnel will contact study participants at 6 weeks, 3 months, 6 months, 9 months, and 37 12 months after their fracture. Our primary outcome will be surgical site infection (SSI) and it will 38 be assessed at 30 days (superficial infections) and at 90 days (deep and organ space infections) 39 after definitive fracture management surgery. The secondary outcome will be occurrence of an 40 unplanned fracture-related reoperation within 12 months of the fracture. Additional time points 41 will be used for our planned sensitivity analyses. 42 43 44

46

50

52

53

54

55

56

57

58

59

60

61

62

63

64

65

66

67

#### 3.0 STATISTICAL PRINCIPLES

#### 3.1 Confidence Intervals and P-Values

All statistical tests will be two-sided and performed using a 5% significance level. We will report all confidence intervals as 95% and two-sided. All results will be expressed as odds ratios produced by analyses described in section 5.2. Interaction p-values will be provided for the subgroup

analyses. We will not adjust for multiple testing, and all sensitivity analyses and secondary results

will be interpreted as exploratory.

#### 3.2 Adherence and Protocol Deviations

in its definition. We will report adherence as the number and percentage of participants who received the allocated intervention at their definitive fracture management surgery. If the participant has multiple open fractures and received the non-allocated treatment at the definitive fracture management surgery for any of their open fractures, we will consider them non-adherent.

Adherence will be assessed at the definitive fracture surgery for each participant and will be binary

We will also tabulate the reasons for non-adherence. The adherence percentages and reasons for

non-adherence will be reported by treatment arm.

Our rationale for defining adherence based solely on the antiseptic solution used during the definitive fracture management surgery is two-fold. 1) The definitive fracture management surgery involves the final implantation of the surgical fixation hardware, when it is most susceptible to bacterial contamination and biofilm development. 2) Any open fracture surgeries prior to the definitive fracture management surgery are staged procedures to remove gross contamination, temporarily stabilize fractures in multi-trauma patients, and minimize evolving soft tissue injuries.

Temporally these procedures occur prior to the surgery of interest for the trial's objectives, and if
bacterial contamination had occurred in one of the proceeding procedures, the repeat surgical
debridement and perioperative antibiotics would reduce the likelihood of persistent occult
infection occurring prior to the definitive fracture surgery.

72

73

#### 3.3 Analysis Populations

- 74 *Intention-to-Treat:* Our primary analysis will use the intention-to-treat approach and will include all enrolled participants in the treatment groups to which their cluster was allocated at the time of
- 76 their first fracture management surgery.

77

78

- As-Treated: One of our sensitivity analyses will be performed on an as-treated population (see
- 79 Section 5.4). The as-treated population will include participants from the intention-to-treat
- 80 population but classified based on the intervention received at their definitive fracture management
- 81 surgery. Participants who do not receive one of the two study interventions will be excluded from
- this analysis. This approach for defining the as-treated treatment groups is a simpler adaptation of
- what was initially proposed in the protocol. This final approach was selected to be consistent with
- 84 the classification of adherence outlined above.

85

#### 4.0 TRIAL POPULATION

## 4.1 Cluster Screening and Eligibility

Prior to commencing the trial, the investigators solicited orthopaedic surgery practices treating open fracture patients in hospitals in the United States and Canada to participate in the trial. All potential clusters completed a feasibility questionnaire prior to initiating start-up activities. To be included in the trial, each cluster had to demonstrate: 1) adequate research personnel infrastructure to manage the study, 2) adequate fracture patient volume to complete enrolment within the study timeline, 3) a commitment from all surgeons to adhere to the assigned interventions, and 4) the ability to procure both study interventions. All hospitals started with a run-in phase of at least 1 month to demonstrate that they could adhere to the trial protocol prior to commencing the study.

We will report the number of clusters (orthopaedic practices) screened, included, and excluded in a flow diagram. The number of clusters excluded by reason has been reported previously. <sup>13</sup> Cluster randomization allocation will be included in the flow diagram, and adherence with treatment allocation during the run-in period by cluster will be summarized using percentages.

## 4.2 Patient Screening and Eligibility

All patients 18 years of age or older who present to a recruiting hospital for treatment of an open fracture(s) of the appendicular skeleton will be screened by a research staff member for participation within 3 weeks of their fracture. Eligible patients must receive surgical debridement of their open fracture wound(s) within 72 hours of their injury, and the open fracture(s) must be managed definitively with a surgical implant (e.g., internal fixation, external fixation, joint prosthesis, etc.). Written informed consent is required for study enrollment to permit the clinical

follow-up of study participants. However, our institutional review board did not require informed consent to occur prior to the study treatment, given the urgent nature of the surgery and the predetermination of the two commonly used interventions with cluster-crossover design. The patients, treating clinicians, and research team members at the participating sites are unmasked to the treatment allocation.

The number of patients screened, included, and excluded will be presented in a flow diagram (**Figure 1**). The figure will consist of the number of patients who were eligible, ineligible, and enrolled. In addition, the number of patients excluded by reason will be summarized. We will also list the number of participants who were enrolled and subsequently deemed ineligible by the Central Adjudication Committee by treatment group and overall. Participants deemed ineligible by a central adjudication committee blinded to the treatment will not be included in any analysis, as per the guidance of Fergusson et al.<sup>14</sup>

## 4.3 Participant Withdrawal

The level of withdrawal will be tabulated and classified as "withdrawal of consent" or "lost to follow-up". Participant deaths will also be tabulated.

#### 4.4 Participant Follow-Up

We will report the number of participants who complete follow-up at 3 months after definitive fracture management surgery and 12 months after their fracture, stratified by treatment allocation.

#### 4.5 Cluster Characteristics

Specific details on characteristics of participating clusters, orthopaedic characteristics, and surgical infection prevention information in the PREPARE Open trial have been previously published.<sup>13</sup>

136

137

138

139

140

141

142

143

144

145

146

147

148

149

150

151

152

153

154

133

134

135

### 4.6 Participant Demographics, Fracture Characteristics, and Descriptions of Surgical and

#### **Perioperative Care**

We will describe the study population with respect to age, sex, race or ethnicity, body mass index, diabetes status, smoking status, Injury Severity Score, the American Society of Anesthesiologists Physical Status Classification System, the number of included open fractures per participant, the severity of the open fracture according to the Gustilo-Anderson classification, <sup>7</sup> the location of the fracture, level of wound contamination using the OTA-OFC classification,<sup>8</sup> the use of temporary fracture stabilization, the number of planned surgeries, the duration of perioperative antibiotic administration, and the method of wound closure (Tables 1 and 2). Categorical data will be summarised by counts with percentages. Age will be summarised as a mean with standard deviation. We will report the Injury Severity Score as a median with an interquartile range. The duration of systemic perioperative antibiotics will be summarised in days and reported as a median with interquartile range. Body mass index (BMI) will be reported in kg/m<sup>2</sup> and subcategorized as underweight (BMI  $\leq$  18.5), normal weight (18.5 – 24.9), overweight (25 – 29.9), and obese (BMI > 30). Additional patient characteristics may be reported as supplemental information. All reporting will be stratified by treatment groups. We will not statistically test for differences in baseline characteristics between treatment groups; however, the clinical importance of any imbalance will be noted.

#### 5.0 ANALYSIS

#### **5.1 Outcome Definitions**

Primary Outcome

Our primary outcome is SSI guided by the Centers for Disease Control and Prevention's (CDC) National Healthcare Safety Network reporting criteria (2017). The SSI surveillance period for all participants, including participants with multiple planned fracture surgeries, will end 30 days after definitive fracture management surgery for superficial SSI and 90 days after definitive fracture management surgery for deep incisional or organ/space SSI. We will also separately report but not statistically test the occurrence of each type of SSI (superficial incisional infections by 30 days, deep incisional infections by 90 days, and organ/space infections by 90 days) by treatment arm. If multiple tissue levels are involved in the infection, the type of SSI will be defined by the deepest tissue layer involved during the surveillance period. Therefore, only one type of SSI per participant will be reported.

CDC National Healthcare Safety Network Surgical Site Infection Reporting Criteria (2017)

| CDC Nation | ai Healthcare Safety Network Surgical Site Infection Reporting Criteria (2017) |
|---|---|
| Outcome | Description |
| Superficial | Date of event for infection may occur from the date of fracture to 30 days after the definitive |
| Incisional | fracture management surgery |
| SSI | AND |
| | involves only skin and subcutaneous tissue of the incision |
| | AND |
| | patient has at least one of the following: |
| | a. purulent drainage from the superficial incision. |
| | <ul> <li>b. organisms identified from an aseptically obtained specimen from the superficial incision or subcutaneous tissue by a culture or non-culture based microbiologic testing method which is performed for purposes of clinical diagnosis or treatment (e.g., not Active Surveillance Culture/Testing [ASC/AST]).</li> <li>c. superficial incision that is deliberately opened by a surgeon, attending physician or other designee and culture or non-culture-based testing is not performed.</li> </ul> |
| | AND |
| | patient has at least one of the following signs or symptoms: pain or tenderness; localized swelling; erythema; or heat. |
| | <ul> <li>d. diagnosis of a superficial incisional SSI by the surgeon or attending physician<br/>or other designee.</li> </ul> |
| | The following do not qualify as criteria for meeting the definition of superficial SSI: |
| | • Diagnosis/treatment of cellulitis (redness/warmth/swelling), by itself, does not meet criterion "d" for superficial incisional SSI. Conversely, an incision that is draining or that |

| Outcome | Description |
|---|---|
| | has organisms identified by culture or non-culture-based testing is not considered a |
| | cellulitis. |
| | A stitch abscess alone (minimal inflammation and discharge confined to the points of |
| | <ul> <li>suture penetration).</li> <li>A localized stab wound or pin site infection- Such an infection might be considered either</li> </ul> |
| | a skin (SKIN) or soft tissue (ST) infection, depending on its depth, but not an SSI |
| | Note: A laparoscopic trocar site for an operative procedure is not considered a stab wound. |
| | An infected burn wound is classified as BURN and is not an SSI. |
| Deep | The date of event for infection may occur from the date of fracture to 90 days after the definitive |
| Incisional | fracture management surgery |
| SSI | AND |
| | involves deep soft tissues of the incision (e.g., fascial and muscle layers) |
| | AND |
| | patient has at least one of the following: a. purulent drainage from the deep incision. |
| | <ul><li>a. purulent drainage from the deep incision.</li><li>b. a deep incision that spontaneously dehisces, or is deliberately opened or aspirated by a</li></ul> |
| | surgeon, attending physician or other designee, and organism is identified by a culture or |
| | non-culture based microbiologic testing method which is performed for purposes of |
| | clinical diagnosis or treatment (e.g., not Active Surveillance Culture/Testing |
| | [ASC/AST]) or culture or non-culture based microbiologic testing method is not |
| | performed |
| | AND |
| | patient has at least one of the following signs or symptoms: fever (>38°C); localized pain or tenderness. A culture or non-culture-based test that has a negative finding does |
| | not meet this criterion. |
| | c. an abscess or other evidence of infection involving the deep incision that is detected on |
| | gross anatomical or histopathologic exam, or imaging test |
| Organ/Space | Date of event for infection may occur from the date of fracture to 90 days after the definitive |
| SSI | fracture management surgery |
| | AND |
| | infection involves any part of the body deeper than the fascial/muscle layers, that is opened or |
| | manipulated during the operative procedure |
| | AND patient has at least one of the following: |
| | a. purulent drainage from a drain that is placed into the organ/space (e.g., closed |
| | suction drainage system, open drain, T-tube drain, CT guided drainage) |
| | b. organisms are identified from an aseptically obtained fluid or tissue in the |
| | organ/space by a culture or non-culture based microbiologic testing method |
| | which is performed for purposes of clinical diagnosis or treatment (e.g., not |
| | Active Surveillance Culture/Testing [ASC/AST]). |
| | c. an abscess or other evidence of infection involving the organ/space that is |
| | detected on gross anatomical or histopathologic exam, or imaging test evidence |
| | suggestive of infection. AND |
| | meets at least one criterion for a specific organ/space infection site summarized in the |
| | Surveillance Definitions for Specific Types of Infections chapter. 1 |
| *The CDC crite | eria have been modified to include all definitive fracture management surgeries instead of including |

<sup>\*</sup>The CDC criteria have been modified to include all definitive fracture management surgeries instead of including only National Healthcare Safety Network procedures that require infection reporting.

## Secondary Outcome

The secondary outcome is the occurrence of an unplanned fracture-related reoperation within 12 months of the fracture. Unplanned reoperations are a common, patient-important outcome in fracture surgery research that captures severe wound and bone healing complications that may be related to occult infections. <sup>15–17</sup> Our definition includes treatments for infection, wound healing complications, or fracture healing complications such as a delayed union or nonunion. We will also report the occurrence of each type of unplanned reoperation by treatment arm.

## **5.2 Analysis Methods**

We will report the number and percentage of patients who sustain the study outcomes by treatment group. We will evaluate the effect of the preoperative antiseptic solutions on our study outcomes using mixed effects regression models with a binomial distribution to produce treatment effect estimates presented as odds ratios with 95% confidence intervals as recommended. For patients with multiple open fractures, the patient will remain the unit of analysis regardless of whether the study event occurs in one or more of their open fractures. As suggested by Morgan et al. and Hemming et al., we will include time and treatment as fixed effects and use random effects to account for the complex correlation structure. We will consider three correlation structures, in the following sequence: exponential decay, nested exchangeable, and exchangeable. If we experience convergence issues or find insufficient between-period correlation to support an exponential decay or nested exchangeable structure, we will assume an exchangeable correlation structure. If we encounter convergence issues even with this model, a more simplified structure will be considered. The models will also include prespecified covariates prognostic of infection or unplanned reoperation as fixed effects. These covariates are the severity of the open fracture,

location of the fracture, and severity of the wound contamination.<sup>22</sup> The same covariates will be used for all primary and secondary outcomes. This planned analysis is a more complex structure than we proposed in the initial study protocol but represents the most recently recommended statistical techniques for cluster-crossover trial analysis.<sup>19,21,23,24</sup> Estimated within-period intracluster correlation coefficients will also be reported.<sup>25</sup>

Our primary and secondary analyses will use multiple imputations to account for missing data. The multiple imputation analysis will create 100 imputed datasets using multivariate imputation by chained equations and pooled using Rubin's rules for combining.<sup>26</sup> The imputation will be performed separately within each treatment arm.

## 5.3 Subgroup Analyses

To determine treatment effect heterogeneity on the study outcomes, we will use the same analytical approach as specified for the primary and secondary outcomes above but include a treatment by subgroup interaction term in the model. We will report results by the prespecified subgroups, which consists of the severity of the open fracture (Gustilo-Anderson type I or II versus type III), upper extremity versus lower extremity open fractures, and the severity of the wound contamination (none, minimal, or surface contamination versus embedded wound contamination) using a forest plot reporting odds ratios with 95% confidence intervals. These analyses will be approached and reported in accordance with best practices and guidelines for subgroup analyses.<sup>27–31</sup> We will use the criteria suggested by Schandelmaier et al. to guide inferences about the credibility of our subgroup analyses.<sup>31</sup> As participants may have more than one included fracture

221

222

223

224

225

226

227

228

229

230

231

232

233

234

235

236

237

238

239

240

241

242

representing different subgroups, the analyses will be performed by categorizing participants according to the fracture with the most severe injury characteristic for each subgroup. **5.4 Sensitivity Analyses** We will consider four alternative analysis approaches to evaluate the robustness of our findings, including alternative definitions of the primary outcome, an as-treated analysis of the primary and secondary outcomes, a complete case missing data analysis of the primary and secondary outcomes, and a Bayesian analysis of the primary and secondary outcomes. We will also allow for post-hoc sensitivity analysis based on information not anticipated in advance. Alternative Definitions of SSI: To evaluate the robustness of the result, we will consider two alternative exploratory definitions of SSI: 1) using the confirmatory criteria from the consensus definition of Fracture-Related Infection (FRI), and 2) expanding the CDC criteria for all types of SSI to within 1 year of injury.<sup>32</sup> Our adjudication of Fracture-Related Infection is defined by the confirmatory criteria outlined in its 2018 consensus definition.<sup>32</sup> The FRI criteria have been selected as an exploratory outcome because the CDC criteria have been criticized for failing to adequately account for the complexities of infections in traumatic fractures. 33,34 The FRI criteria attempt to improve the ability to detect infections specifically in fracture patients; however, this definition of FRI has not been fully validated or widely adopted. The confirmatory criteria include the presence of one or more of the following signs/symptoms:

- 243 1) Fistula, sinus, or wound breakdown (with communication to the bone or the implant).
  - 2) Purulent drainage from the wound or presence of pus during surgery.
    - 3) Phenotypically indistinguishable pathogens identified by culture from at least two separate deep tissue/implant (including sonication-fluid) specimens taken during an operative intervention. In the case of tissue, multiple specimens (3) should be taken, each with clean instruments (not superficial or sinus tract swabs). In cases of joint effusion arising in a joint adjacent to a fractured bone, fluid samples obtained by sterile puncture may be included as a single sample.
    - 4) Presence of microorganisms in deep tissue taken during an operative intervention, as confirmed by histopathological examination using specific staining techniques for bacteria or fungi.

The second exploratory definition of surgical site infection expands the CDC criteria to a 12-month surveillance period. This outcome will use the same diagnostic CDC reporting criteria for the primary; however, the timeframe for this outcome will be expanded to include all SSIs that occur within 12 months of open fracture. Similar to the rationale for using the FRI outcome and the recommendations for a minimum of 12 months follow-up for orthopaedic fracture outcomes, this expanded timeframe will detect infections that occur beyond the standard CDC surveillance reporting periods. This modification of the CDC reporting periods has been used in previous orthopaedic fracture trials. 15,35

As-Treated Analysis: One of our sensitivity analyses will be performed on an as-treated population.

The as-treated population will include participants from the intention-to-treat population who

received one of the two interventions; however, participants will be classified based on the intervention received at their definitive fracture management surgery. Participants who do not receive one of the study interventions will be removed from this analysis. Similar to the primary analysis, we will use mixed effects regression models with a binomial distribution and the same covariates and correlation structure as the primary model. A more simplified structure will be considered if we encounter convergence issues with this model.

Missing Data: While we anticipate minimal missing outcome data, we will perform a sensitivity analysis on the primary and secondary analyses to explore the impact of missing outcome data. Our sensitivity analysis will be a complete case analysis, including only those patients with a known status of the outcome being analyzed.

Bayesian Analysis: The Bayesian analyses will be performed using four different priors (neutral with moderate strength, neutral flat, optimistic with moderate strength, and pessimistic with moderate strength) defined on a log-odds scale and described below. The neutral priors will be centered on a log odds of 0 (odds ratio of 1). The neutral flat prior will have a standard deviation of 100. The optimistic prior will be centered on the estimated effect size of a 0.62 odds ratio (log odds of -0.48). In contrast, the pessimistic prior is centered on the same effect size but for the alternative treatment. As suggested by Zampieri et al.,<sup>36</sup> the standard deviation of 0.48 was selected for the moderate strength priors as it allows for a 15% probability of the alternative treatment benefit in both the optimistic and pessimistic prior. The prior probability of our neutral prior with a moderate strength distribution implies a 68% chance the estimated effect will be between an odds

ratio of 0.62 and 1.38. The neutral prior with moderate strength will be our preferred prior in this sensitivity analysis.

The modeling for the Bayesian analysis will be consistent with our primary analysis. We will use a mixed effects regression model with a Bernoulli distribution. The model will include time and treatment as fixed effects and use random effects to account for the complex correlation structure. The best fitting correlation structure will be determined using information criteria. If we experience convergence issues with this model structure, we will transition to a less complex model. We will report treatment effects as odds ratios with 95% credible intervals. We will also report the probability of treatment benefits of povidone-iodine, with 50% implying no difference in the probability of benefit between the two treatment groups.

## Priors used in the analysis with their interpretation and a visual depiction.

| Prior | Mean | Standard Deviation | Interpretation | Visualization |
|---|---|---|---|---|
| Neutral<br>with<br>moderate<br>strength | Log(1.00)<br>= 0 | 0.48 | "There is no strong information to suggest the intervention is good or bad in this study population, but we think extreme effect sizes are very unlikely." | Favors Povidone-Iodine Favors Chlorhexidine 0.8 0.8 0.0 0.22 0.62 1.38 Odds Ratio |
| Neutral flat | Log(1.00)<br>= 0 | 100 | "None of the prior<br>research is relevant to<br>this trial, and we<br>cannot rule out<br>extreme effect sizes." | Favors Povidone-Iodine Favors Chlorhexidine 0.4 0.0 0.2 0.82 1.38 0.38 0.48 0.49 0.40 0.40 0.50 |

| Optimistic with moderate strength | Log(0.62)<br>= -0.48 | 0.48 | "We think povidone- iodine is more effective but cannot rule out that chlorhexidine is superior." | Favors Povidone-Iodine Favors Chlorhexidine 0.4 0.0 0.22 0.82 1.38 0.338 Odds Ratio |
|---|---|---|---|---|
| Pessimistic with moderate strength | Log(1.38)<br>= 0.32 | 0.48 | "We think<br>chlorhexidine is more<br>effective but cannot<br>rule out that povidone-<br>iodine is superior." | Favors Povidone-lodine Favors Chlorhexidine 0.4 0.2 0.62 1.38 Odds Ratio |

5.5 Harms

301

302

303

304

305

306

307

308

309

The number and percentage of patients experiencing serious adverse events will be presented by treatment arm. No formal statistical testing will be undertaken.

**5.6 Statistical Software** 

The statistical analyses will be performed with SAS, version 9.4 (SAS Institute, Cary, NC) and R (R Foundation for Statistical Computing, Vienna, Austria).

# 6.0 FIGURES AND TABLES

310

# **Table 1: Baseline characteristics**

| | Iodine Povacrylex in | Chlorhexidine in |
|---|---|---|
| | Alcohol | Alcohol |
| A (GD) | (n= XX participants) | (n= XX participants) |
| Age, years, mean (SD) | | |
| Sex, n (%) | | |
| Female | | |
| Male | | |
| Prefer not to answer | | |
| Race or ethnicity, n (%) | | |
| White | | |
| Black | | |
| Central or South American | | |
| Asian | | |
| Indigenous | | |
| Native Hawaiian or Pacific Islander | | |
| Multiracial | | |
| Prefer not to answer | | |
| Body mass index, kg/m <sup>2</sup> , n (%) | | |
| Underweight (BMI < 18·5) | | |
| Normal weight $(18.5 - 24.9)$ | | |
| Overweight (25 – 29·9) | | |
| Obese (BMI > 30) | | |
| Diabetes, n (%) | | |
| Current smoker, n (%) | | |
| Injury severity score, mean (SD) | | |
| American Society of Anesthesiologist | | |
| Physical Score, n (%) | | |
| Class I or II | | |
| Class III or higher | | |
| Number of included open fractures per | | |
| participant, n (%) | | |
| One | | |
| Two | | |
| Three | | |

315

316 317

318

313 Table 2: Fracture Characteristics and Management

| | Iodine Povacrylex in<br>Alcohol | Chlorhexidine in<br>Alcohol |
|---|---|---|
| | (n= XX fractures) | (n= XX fractures) |
| Severity of open fracture, n (%) | | |
| Gustilo-Anderson type I | | |
| Gustilo-Anderson type II | | |
| Gustilo-Anderson type IIIA | | |
| Gustilo-Anderson type IIIB/IIC | | |
| Location of fracture, n (%) | | |
| Lower extremity or pelvis | | |
| Upper extremity | | |
| Wound contamination, n (%) | | |
| None or minimal contamination | | |
| Surface contamination | | |
| Contaminant embedded in bone or deep soft | | |
| tissue | | |
| Temporary fracture stabilization, n (%) | | |
| Number of planned surgeries, n (%) | | |
| 1 | | |
| 2 | | |
| 3 | | |
| 4 | | |
| 5 or more | | |
| Duration of antibiotic administration (days), | | |
| median (IQR) | | |
| Closure method, n (%)* | | |
| Primary wound closure | | |
| No closure attempted/secondary wound | | |
| healing | | |
| Skin graft | | |
| Local flap | | |
| Free flap *More than one type of closure method may have been not | | |

<sup>\*</sup>More than one type of closure method may have been performed during surgery, but only the most complex method of closure is reported in the table using the following the hierarchy: 1) free flap, 2) local flap, 3) skin graft, 4) no closure attempted/secondary wound healing, 5) primary wound closure

319 **Table 3: Study outcomes** 

| | Iodine Povacrylex in<br>Alcohol (n=XXX)<br>number (%)* | Chlorhexidine in<br>Alcohol (n=XXX)<br>number (%)* | Odds<br>Ratio** | p-value** | Risk Difference** |
|---|---|---|---|---|---|
| Primary outcome | n=XXX | n=XXX | (95% CI) | | (95% CI) |
| Surgical site infection | 11 717171 | 11 747474 | | | |
| Superficial infection | | | | | |
| Deep incisional | | | | | |
| Organ/space infection | | | | | |
| | | | | , | |
| Alternative definitions of surgical site | n=XXX | n=XXX | | | |
| infection | | | | | |
| Any surgical site infection by 365 | | | | | |
| days | | | | | |
| Fracture-related infection by 365 days | | | | | |
| Secondary outcome | n=XXX | n=XXX | | | |
| Unplanned reoperation by 365 days | | | | | |
| Unplanned reoperation for infection | | | | | |
| by 365 days | | | | | |
| Unplanned reoperation for wound | | | | | |
| healing complications by 365 days | | | | | |
| Unplanned reoperation to promote | | | | | |
| fracture healing by 365 days | | | | | |

CI = Confidence Interval

<sup>320</sup> 321 322 \*Percentages based on complete case description
\*\*Missing outcome data were imputed using multiple imputations 323



## Figure 2. Forest plot of subgroup analyses



## LIST OF ABBREVIATIONS

4 5

3

ASC/AST Active surveillance culture/testing

PREPARE A Pragmatic Randomized trial Evaluating Pre-operative Alcohol

skin solutions in FRactured Extremities

BMI Body mass index

CDC Centers for Disease Control

FRI Fracture-related infection

OTA-OFC Orthopaedic Trauma Association open fracture classification

ST Soft tissue

SSI Surgical site infection

6

7

9 **DECLARATIONS** 10 **Ethics Approval and Consent to Participate** 11 12 Ethics approval has been obtained from the Hamilton Integrated Research Ethics Board for the 13 Methods Center (#4336), the Advarra Central Institutional Review Board (formerly Chesapeake 14 Institutional Review Board) (#Pro00023709), and each clinical site's local institutional review 15 board or research ethics board, if they are not using the central institutional review board. Written 16 informed consent has been obtained for study participation. 17 18 **Consent for Publication** 19 Not applicable 20 21 **Availability of Data and Materials** 22 The datasets generated and/or analyzed during the current study are not publicly available due to 23 the trial still being ongoing, but will be available from the corresponding author on reasonable 24 request. 25 26 **Competing Interests** 27 Dr. Slobogean reports editorial or governing board for the Journal of Orthopaedic Trauma, board 28 or committee member for the Orthopaedic Trauma Association, paid consultant for Smith & 29 Nephew, and paid consultant for Zimmer, all outside the submitted work. Dr. Sprague reports 30 board or committee member for Orthopaedic Trauma Association, employment from Global 31 Research Solutions Inc. and consultant fees from the University of Sherbrooke and Platform Life 32 Sciences, all outside the submitted work. Dr. Bhandari reports paid consultant from AgNovos

- Healthcare, research support from the Canadian Institutes of Health Research (CIHR), board or committee member for the International Society of Orthopaedic Surgery and Traumatology (SICOT), research support from the National Institutes of Health (NIAMS & NICHD), research support from Physicians' Services Incorporated, paid consultant for Sanofi-Aventis, paid consultant for Smith & Nephew, and research support from the U.S. Department of Defense, all outside the submitted work. Dr. O'Hara reports stock or stock options from Arbutus Medical Inc,
- 40

39

- 41 Funding
- The PREPARE trial is funded by the Patient-Centered Outcomes Research Institute (PCS-1609-
- 43 36512) and the Canadian Institutes of Health Research (Foundation Grant).

all outside the submitted work. All other authors have nothing to report.

#### 45 Authors' Contributions

- 46 All authors have been major contributors in writing the statistical analysis plan. All authors have
- 47 read and approved the statistical analysis plan.
- 48
- 49 Acknowledgements

**PREP-IT Investigators** 

- 50 51
- 52 Executive Committee: Gerard P. Slobogean (Principal Investigator, University of Maryland
- 53 School of Medicine, Baltimore, MD); Sheila Sprague (Principal Investigator, McMaster
- 54 University, Hamilton, ON); Jeffrey L. Wells (Patient Representative, Trauma Survivors Network,
- Falls Church, VA); Mohit Bhandari (Principal Investigator, McMaster University, Hamilton, ON)
- 56
- 57 Steering Committee: Gerard P. Slobogean (Co-Chair, University of Maryland School of
- Medicine, Baltimore, MD); Mohit Bhandari (Co-Chair, McMaster University, Hamilton, ON);
- 59 Sheila Sprague (Principal Investigator, McMaster University, Hamilton, ON); Anthony D. Harris
- 60 (University of Maryland School of Medicine, Baltimore, MD); C. Daniel Mullins (University of
- 61 Maryland School of Medicine, Baltimore, MD); Lehana Thabane (McMaster University,

Hamilton, ON); Jeffrey L. Wells (Trauma Survivors Network, Falls Church, VA); Amber Wood (Association of periOperative Registered Nurses, Denver, CO)

Adjudication Committee: Gregory J. Della Rocca (Chair, University of Missouri, Columbia, MO); Anthony D. Harris (University of Maryland School of Medicine, Baltimore, MD); Joan N. Hebden (University of Maryland School of Medicine, Baltimore, MD); Kyle J. Jeray (Prisma Health - Upstate, Greenville, SC); Lucas S. Marchand (University of Utah, Salt Lake City, UT); Lyndsay M. O'Hara (University of Maryland School of Medicine, Baltimore, MD); Robert D. Zura (LSU Health, New Orleans, LA); Christopher Lee (University of California, Los Angeles, CA); Joseph T. Patterson (University of Southern California, Los Angeles, CA)

**Data and Safety Monitoring Committee:** Michael J. Gardner (Chair, Stanford University School of Medicine, Palo Alto, CA); Jenna Blasman (Patient Representative, Kitchener, ON); Jonah Davies (University of Washington, Seattle, WA); Stephen Liang (Washington University, St. Louis, MO); Monica Taljaard (Ottawa Hospital Research Institute, Ottawa, ON)

**Research Methodology Core:** PJ Devereaux (McMaster University, Hamilton, ON); Gordon Guyatt (McMaster University, Hamilton, ON); Lehana Thabane (McMaster University, Hamilton, ON); Diane Heels-Ansdell (McMaster University, Hamilton, ON)

 Patient Centred Outcomes Core: Debra Marvel (Patient Representative, Baltimore, MD); Jana E. Palmer (Patient Representative, Baltimore, MD); Jeffrey L. Wells (Patient Representative, Trauma Survivors Network, Falls Church, VA); Jeff Friedrich (Editor, Slate Magazine, Washington, DC); C. Daniel Mullins (University of Maryland School of Medicine, Baltimore, MD); Nathan N. O'Hara (University of Maryland School of Medicine, Baltimore, MD); Frances Grissom (Trauma Survivor Network, Baltimore, MD)

**Orthopaedic Surgery Core:** Gregory J. Della Rocca (University of Missouri, Columbia, MO); I. Leah Gitajn (Dartmouth University, Hanover, NH); Kyle J. Jeray (Prisma Health - Upstate, Greenville, SC); Saam Morshed (San Francisco General Hospital, San Francisco, CA); Robert V. O'Toole (University of Maryland School of Medicine, Baltimore, MD); Bradley Petrisor (Hamilton Health Sciences, Hamilton, ON)

Operating Room Core: Franca Mossuto (Hamilton Health Sciences, Hamilton, ON)
Infectious Disease Core: Anthony D. Harris (University of Maryland School of Medicine, Baltimore, MD); Manjari G. Joshi (University of Maryland School of Medicine, Baltimore, MD)

**Military Core:** Jean-Claude G. D'Alleyrand (Walter Reed National Military Medical Center, 100 Bethesda, MD); Justin Fowler (United States Army, USA); Jessica C. Rivera (San Antonio 101 Military Medical Center, San Antonio, TX); Max Talbot (Canadian Armed Forces, Montreal, QC)

- McMaster University Methods Center (Hamilton, ON): Sheila Sprague (Principal Investigator);
   Mohit Bhandari (Principal Investigator); David Pogorzelski (Research Coordinator); Shannon
- Dodds (Research Coordinator); Silvia Li (Research Coordinator); Gina Del Fabbro (Research
- 106 Assistant); Olivia Paige Szasz (Research Assistant); Diane Heels-Ansdell (Statistician); Paula

- 107 McKay (Manager); Alexandra Minea (Research Coordinator); Kevin Murphy (Research
- 108 Assistant); Sofia Bzovsky (Statistical Analyst)
- 110 University of Maryland School of Medicine Administrative Center (Baltimore, MD): Gerard
- P. Slobogean (Principal Investigator); Nathan N. O'Hara (Manager); Andrea L. Howe (Project
- Manager); Haley Demyanovich (Project Manager), Wayne Hoskins (Co-Investigator)
- 114 University of Maryland School of Pharmacy, The PATIENTS Program (Baltimore, MD): C.
- Daniel Mullins (Executive Director); Michelle Medeiros (Director of Research); Genevieve Polk
- 116 (Assistant Director, Dissemination and Research); Eric Kettering (Senior Instructional Technology
- and Dissemination Specialist); Nirmen Mahal (Program Specialist)
- 119 **PREP-IT Clinical Sites:**

113

118

126

131

143

148

- 120 Lead Clinical Site (Aqueous-PREP and PREPARE):
- 121 University of Maryland School of Medicine, R Adams Cowley Shock Trauma Center,
- Baltimore, MD: Robert V. O'Toole, Jean-Claude G. D'Alleyrand, Andrew Eglseder, Aaron
- 123 Johnson, Christopher Langhammer, Christopher Lebrun, Jason Nascone, Raymond Pensy,
- 124 Andrew Pollak, Marcus Sciadini, Gerard P. Slobogean, Yasmin Degani, Haley K. Demyanovich,
- 125 Andrea L. Howe, Nathan N. O'Hara, Heather Phipps, Eric Hempen
- 127 Aqueous-PREP and PREPARE:
- Hamilton Health Sciences General Site, Hamilton, ON: Bradley Petrisor, Herman Johal, Bill
- Ristevski, Dale Williams, Matthew Denkers, Krishan Rajaratnam, Jamal Al-Asiri, Jodi L. Gallant,
- 130 Kaitlyn Pusztai, Sarah MacRae, Sara Renaud.
- 132 **Prisma Health Upstate, Greenville, SC**: Kyle J. Jeray, John D. Adams, Michael L. Beckish,
- 133 Christopher C. Bray, Timothy R. Brown, Andrew W. Cross, Timothy Dew, Gregory K. Faucher,
- Richard W. Gurich Jr, David E. Lazarus, S. John Millon, M. Christian Moody, M. Jason Palmer,
- Scott E. Porter, Thomas M. Schaller, Michael S. Sridhar, John L. Sanders, L. Edwin Rudisill, Jr.
- Michael J. Garitty, Andrew S. Poole, Michael L. Sims, Clark M. Walker, Robert Carlisle, Erin A.
- Hofer, Brandon Huggins, Michael Hunter, William Marshall, Shea B. Ray, Cory Smith, Kyle M.
- Altman, Erin Pichiotino, Julia C. Quirion, Markus F. Loeffler, Erin R. Pichiotino, Austin A. Cole,
- Ethan J. Maltz, Wesley Parker, T. Bennett Ramsey, Alex Burnikel, Michael Colello, Russell
- 140 Stewart, Jeremy Wise, Matthew Anderson, Joshua Eskew, Benjamin Judkins, James M. Miller,
- 141 Stephanie L. Tanner, Rebecca G. Snider, Christine E. Townsend, Kayla H. Pham, Abigail Martin,
- Emily Robertson, Emily Bray, J. Wilson Sykes, Krystina Yoder, Kelsey Conner, Harper Abbott
- 144 IU Health Methodist Hospital, Indianapolis, IN: Roman M. Natoli, Todd O. McKinley, Walter
- W. Virkus, Anthony T. Sorkin, Jan P. Szatkowski, Brian H. Mullis, Yohan Jang, Luke A. Lopas,
- Lauren C. Hill, Courteney L. Fentz, Maricela M. Diaz, Krista Brown, Katelyn M. Garst, Emma
- 147 W. Denari
- 149 San Antonio Military Medical Center, San Antonio, TX: Patrick Osborn, Justin Fowler, Sarah
- N. Pierrie, Bradley Kessler, Maria Herrera

- 152 University of California, San Francisco, San Francisco, CA: Saam Morshed, Theodore
- 153 Miclau, Meir T. Marmor, Amir Matityahu, R. Trigg McClellan, David Shearer, Paul Toogood,
- Anthony Ding, Jothi Murali, Ashraf El Naga, Jennifer Tangtiphaiboontana, Tigist Belaye, Eleni
- 155 Berhaneselase, Dmitry Pokhvashchev
- 156
- 157 Aqueous-PREP:
- Vanderbilt Medical Center, Nashville, TN: William T. Obremskey, Amir Alex Jahangir, Manish
- 159 Sethi, Robert Boyce, Daniel J. Stinner, Phillip P. Mitchell, Karen Trochez, Elsa Rodriguez, Charles
- 160 Pritchett, Natalie Hogan, A. Fidel Moreno

- 162 University of Florida, Gainesville, FL: Jennifer E. Hagen, Matthew Patrick, Richard Vlasak,
- 163 Thomas Krupko, Michael Talerico, Marybeth Horodyski, Marissa Pazik, Elizabeth Lossada-Soto

164

- McGovern Medical School at UTHealth Houston, Houston, TX: Joshua L. Gary, Stephen J.
- Warner, John W. Munz, Andrew M. Choo, Timothy S. Achor, Milton L. "Chip" Routt, Michael
- 167 Kutzler, Sterling Boutte, Ryan J. Warth

168

- Wright State University, Dayton, OH: Michael J. Prayson, Indresh Venkatarayappa, Brandon
- Horne, Jennifer Jerele, Linda Clark

171

- 172 Banner University Medical Center Tucson, Tucson, AZ: Christina Boulton, Jason Lowe,
- John T. Ruth, Brad Askam, Andrea Seach, Alejandro Cruz, Breanna Featherston, Robin Carlson,
- 174 Iliana Romero, Isaac Zarif

175

- 176 The CORE Institute, Phoenix, AZ: Niloofar Dehghan, Michael McKee, Clifford B. Jones, Debra
- 177 L. Sietsema, Alyse Williams, Tayler Dykes

178

- 179 Vall d'Hebron University Hospital, Barcelona, Spain: Ernesto Guerra-Farfan, Jordi Tomas-
- Hernandez, Jordi Teixidor-Serra, Vicente Molero-Garcia, Jordi Selga-Marsa, Juan Antonio
- Porcel-Vazquez, Jose Vicente Andres-Peiro, Ignacio Esteban-Feliu, Nuria Vidal-Tarrason, Jordi
- 182 Serracanta, Jorge Nuñez-Camarena, Maria del Mar Villar-Casares, Jaume Mestre-Torres, Pilar
- 183 Lalueza-Broto, Felipe Moreira-Borim, Yaiza Garcia-Sanchez

184

- 185 Hospital Universitari Parc Tauli, Barcelona, Spain: Francesc Marcano-Fernández, Laia
- Martínez-Carreres, David Martí-Garín, Jorge Serrano-Sanz, Joel Sánchez-Fernández, Matsuyama
- 187 Sanz-Molero, Alejandro Carballo, Xavier Pelfort, Francesc Acerboni-Flores, Anna Alavedra-
- 188 Massana, Neus Anglada-Torres, Alexandre Berenguer, Jaume Cámara-Cabrera, Ariadna
- Caparros-García, Ferran Fillat-Gomà, Ruben Fuentes-López, Ramona Garcia-Rodriguez, Nuria
- 190 Gimeno-Calavia, Marta Martínez-Álvarez, Patricia Martínez-Grau, Raúl Pellejero-García, Ona
- 191 Ràfols-Perramon, Juan Manuel Peñalver, Mònica Salomó Domènech, Albert Soler-Cano, Aldo
- 192 Velasco-Barrera, Christian Yela-Verdú, Mercedes Bueno-Ruiz, Estrella Sánchez-Palomino, Vito
- 193 Andriola, Matilde Molina-Corbacho, Yeray Maldonado-Sotoca, Alfons Gasset-Teixidor, Jorge
- 194 Blasco-Moreu, Núria Fernández-Poch, Josep Rodoreda-Puigdemasa, Arnau Verdaguer-Figuerola,
- 195 Heber Enrique Cueva-Sevieri, Santiago Garcia-Gimenez

196

197 PREPARE:

- 198 FRASER HEALTH AUTHORITY/Royal Columbian Hospital, New Westminster, BC:
- Darius G. Viskontas, Kelly L. Apostle, Dory S. Boyer, Farhad O. Moola, Bertrand H. Perey,
- Trevor B. Stone, H. Michael Lemke, Ella Spicer, Kyrsten Payne
- 201
- 202 Inova Fairfax Medical Campus, Falls Church, VA: Robert A. Hymes, Cary C. Schwartzbach,
- Jeff E. Schulman, A. Stephen Malekzadeh, Michael A. Holzman, Greg E. Gaski, Jonathan Wills,
- 204
- Wake Forest Baptist Health, Winston-Salem, NC: Holly Pilson, Eben A. Carroll, Jason J.
- Halvorson, Sharon Babcock, J. Brett Goodman, Martha B. Holden, Wendy Williams, Taylor Hill,
- 207 Ariel Brotherton
- 208
- 209 MetroHealth Medical Center, Cleveland, OH: Nicholas M. Romeo, Heather A. Vallier, Anna
- 210 Vergon
- 211
- 212 University of Utah, Salt Lake City, Utah: Thomas F. Higgins, Justin M. Haller, David L.
- 213 Rothberg, Lucas S. Marchand, Zachary M. Olsen, Abby V. McGowan, Sophia Hill, Morgan K.
- 214 Dauk
- 215
- 216 University of Mississippi Medical Center, Jackson, MS: Patrick F. Bergin, George V. Russell,
- 217 Matthew L. Graves, John Morellato, Sheketha L. McGee, Eldrin L. Bhanat, Ugur Yener, Rajinder
- 218 Khanna, Priyanka Nehete
- 219
- 220 Sanford Health, Sioux Falls, SD: David Potter, Robert VanDemark III, Kyle Seabold, Nicholas
- 221 Staudenmier
- 222
- 223 Dartmouth-Hitchcock Medical Center, Lebanon, NH: I. Leah Gitajn, Marcus Coe, Kevin
- Dwyer, Devin S. Mullin, Theresa A. Chockbengboun, Peter A. DePalo Sr.
- 225
- 226 Carolinas Medical Center, Atrium Health Musculoskeletal Institute, Charlotte, NC: Kevin
- 227 Phelps, Michael Bosse, Madhay Karunakar, Laurence Kempton, Stephen Sims, Joseph Hsu,
- 228 Rachel Seymour, Christine Churchill, Ada Mayfield, Juliette Sweeney
- 229
- 230 University of Maryland, Capital Region Health: Largo, MD: Todd Jaeblon, Robert Beer, Haley
- 231 K. Demyanovich, Brent Bauer, Sean Meredith, Sneh Talwar
- 232
- 233 University of Wisconsin Madison, Madison, WI: Christopher M. Domes
- 234
- Duke University Hospital, Durham, NC: Mark J. Gage, Rachel M. Reilly, Ariana Paniagua,
- JaNell Dupree
- 237
- 238 Brigham Women's Hospital, Boston, MA: Michael J. Weaver, Arvind G. von Keudell, Abigail
- E. Sagona
- 240
- 241 University of Pennsylvania, Philadelphia, PA: Samir Mehta, Derek Donegan, Annamarie
- 242 Horan, Mary Dooley
- 243

244 Massachusetts General Hospital, Boston, MA: Marilyn Heng, Mitchel B. Harris, David W. 245 Lhowe, John G. Esposito, Ahmad Alnasser 246 247 Bryan Medical Center, Lincoln, Nebraska: Steven F. Shannon, Alesha N. Scott, Bobbi Clinch, 248 Becky Weber 249 250 University of Cincinnati, Cincinnati, OH: Michael J. Beltran, Michael T. Archdeacon, Henry 251 Claude Sagi, John D. Wyrick, Theodore Toan Le, Richard T. Laughlin, Cameron G. Thomson, 252 Kimberly Hasselfeld 253 254 Cedars-Sinai Medical Center, Los Angeles, CA: Carol A. Lin, Mark S. Vrahas, Charles N. 255 Moon, Milton T. Little, Geoffrey S. Marecek, Denice M. Dubuclet 256 257 University of California, Irvine, Orange, CA: John A. Scolaro, James R. Learned, Philip K. Lim, Susan Demas, Arya Amirhekmat, Yan Marco Dela Cruz 258 259 260

- 261 REFERENCES
- 262 1. Centers for Disease Control and Prevention (CDC). Surgical Site Infection (SSI) Event.;
- 263 2017.
- Darouiche RO, Wall MJ, Itani KMF, et al. Chlorhexidine-Alcohol versus Povidone-Iodine for Surgical-Site Antisepsis. *N Engl J Med*. 2010;362(1):18-26.
- Tuuli MG, Liu J, Stout MJ, et al. A Randomized Trial Comparing Skin Antiseptic Agents at Cesarean Delivery. *N Engl J Med*. 2016;374(7):647-655.
- Swenson BR, Sawyer RG. Importance of alcohol in skin preparation protocols. *Infect Control Hosp Epidemiol*. 2010;31(9):977.
- Swenson BR, Hedrick TL, Metzger R, Bonatti H, Pruett TL, Sawyer RG. Effects of
   preoperative skin preparation on postoperative wound infection rates: a prospective study of
   3 skin preparation protocols. *Infect Control Hosp Epidemiol*. 2009;30(10):964-971.
- FLOW Investigators, Bhandari M, Jeray KJ, et al. A Trial of Wound Irrigation in the Initial
   Management of Open Fracture Wounds. N Engl J Med. 2015;373(27):2629-2641.
   doi:10.1056/NEJMoa1508502
- Gustilo RB, Anderson JT. Prevention of infection in the treatment of one thousand and twenty-five open fractures of long bones: retrospective and prospective analyses. *J Bone Joint Surg Am.* 1976;58(4):453-458.
- Orthopaedic Trauma Association: Open Fracture Study Group. A new classification scheme for open fractures. *J Orthop Trauma*. 2010;24(8):457-464.
   doi:10.1097/BOT.0b013e3181c7cb6b
- 9. McDonnell G, Russell AD. Antiseptics and disinfectants: activity, action, and resistance. *Clin Microbiol Rev.* 1999;12(1):147-179. doi:10.1128/CMR.12.1.147
- 284 10. Kunisada T, Yamada K, Oda S, Hara O. Investigation on the efficacy of povidone-iodine
   285 against antiseptic-resistant species. *Dermatol Basel Switz*. 1997;195 Suppl 2:14-18.
   286 doi:10.1159/000246025
- 287 11. Gamble C, Krishan A, Stocken D, et al. Guidelines for the Content of Statistical Analysis Plans in Clinical Trials. *JAMA*. 2017;318(23):2337. doi:10.1001/jama.2017.18556
- 289 12. Dwan K, Li T, Altman DG, Elbourne D. CONSORT 2010 statement: extension to randomised crossover trials. *BMJ*. Published online July 31, 2019:14378.
  291 doi:10.1136/bmj.14378
- 292 13. Sprague S, Scott T, Dodds S, et al. Cluster identification, selection, and description in cluster randomized crossover trials: the PREP-IT trials. *Trials*. 2020;21(1):712.

- 294 14. Fergusson D, Aaron SD, Guyatt G, Hébert P. Post-randomisation exclusions: the intention
- to treat principle and excluding patients from analysis. *BMJ*. 2002;325(7365):652-654.
- 296 doi:10.1136/bmj.325.7365.652
- 15. FLOW Investigators, Bhandari M, Jeray KJ, et al. A Trial of Wound Irrigation in the Initial Management of Open Fracture Wounds. *N Engl J Med*. 2015;373(27):2629-2641.
- 299 16. FAITH Investigators. Fracture fixation in the operative management of hip fractures 300 (FAITH): an international, multicentre, randomised controlled trial. *Lancet Lond Engl.*
- 301 2017;389(10078):1519-1527. doi:10.1016/S0140-6736(17)30066-1
- 302 17. HEALTH Investigators, Bhandari M, Einhorn TA, et al. Total Hip Arthroplasty or
- Hemiarthroplasty for Hip Fracture. *N Engl J Med*. 2019;381(23):2199-2208.
- 304 doi:10.1056/NEJMoa1906190
- 305 18. the CONSORT Group, Schulz KF, Altman DG, Moher D. CONSORT 2010 Statement:
- 306 updated guidelines for reporting parallel group randomised trials. *Trials*. 2010;11(1):32.
- 307 doi:10.1186/1745-6215-11-32
- 308 19. Morgan KE, Forbes AB, Keogh RH, Jairath V, Kahan BC. Choosing appropriate analysis
- methods for cluster randomised cross-over trials with a binary outcome: K. E. MORGAN
- 310 ET AL. Stat Med. 2017;36(2):318-333. doi:10.1002/sim.7137
- 311 20. Hemming K, Kasza J, Hooper R, Forbes A, Taljaard M. A tutorial on sample size
- 312 calculation for multiple-period cluster randomized parallel, cross-over and stepped-wedge
- trials using the Shiny CRT Calculator. *Int J Epidemiol*. 2020;49(3):979-995.
- 314 doi:10.1093/ije/dyz237
- 315 21. Hemming K, Taljaard M, Weijer C, Forbes AB. Use of multiple period, cluster randomised,
- crossover trial designs for comparative effectiveness research. *BMJ*. Published online
- November 4, 2020:m3800. doi:10.1136/bmj.m3800
- 318 22. Wise BT, Connelly D, Rocca M, et al. A Predictive Score for Determining Risk of Surgical
- 319 Site Infection After Orthopaedic Trauma Surgery. *J Orthop Trauma*. 2019;33(10):506-513.
- 320 doi:10.1097/BOT.000000000001513
- 321 23. Thompson DD, Lingsma HF, Whiteley WN, Murray GD, Steyerberg EW. Covariate
- adjustment had similar benefits in small and large randomized controlled trials. *J Clin*
- 323 Epidemiol. 2015;68(9):1068-1075. doi:10.1016/j.jclinepi.2014.11.001
- 324 24. Program of Randomized Trials to Evaluate Pre-operative Antiseptic Skin Solutions in
- Orthopaedic Trauma (PREP-IT) Investigators, Slobogean GP, Sprague S, et al.
- 326 Effectiveness of Iodophor vs Chlorhexidine Solutions for Surgical Site Infections and
- 327 Unplanned Reoperations for Patients Who Underwent Fracture Repair: The PREP-IT
- 328 Master Protocol. *JAMA Netw Open*. 2020;3(4):e202215.

- 329 25. Campbell MK, Piaggio G, Elbourne DR, Altman DG, CONSORT Group. Consort 2010
- 330 statement: extension to cluster randomised trials. BMJ. 2012;345:e5661.
- 331 doi:10.1136/bmj.e5661
- 332 26. Rubin DB. Multiple imputation for survey nonresponse. Published online 1987.
- 333 27. Wang R, Lagakos SW, Ware JH, Hunter DJ, Drazen JM. Statistics in medicine--reporting of subgroup analyses in clinical trials. N Engl J Med. 2007;357(21):2189-2194. 334
- 335 28. Sun X, Ioannidis JPA, Agoritsas T, Alba AC, Guyatt G. How to use a subgroup analysis:
- users' guide to the medical literature. JAMA. 2014;311(4):405-411. 336
- 337 29. Sun X. Briel M. Walter SD. Guyatt GH. Is a subgroup effect believable? Updating criteria 338 to evaluate the credibility of subgroup analyses. *BMJ*. 2010;340:c117.
- 339 30. Sun X, Briel M, Busse JW, et al. Subgroup Analysis of Trials Is Rarely Easy (SATIRE): a 340 study protocol for a systematic review to characterize the analysis, reporting, and claim of
- 341 subgroup effects in randomized trials. *Trials*. 2009;10:101.
- 342 Schandelmaier S, Briel M, Varadhan R, et al. Development of the Instrument to assess the
- 343 Credibility of Effect Modification Analyses (ICEMAN) in randomized controlled trials and
- 344 meta-analyses. CMAJ Can Med Assoc J J Assoc Medicale Can. 2020;192(32):E901-E906.
- 345 doi:10.1503/cmaj.200077
- 346 32. Metsemakers Wi, Morgenstern M, McNally MA, et al. Fracture-related infection: A
- 347 consensus on definition from an international expert group. *Injury*. 2018;49(3):505-510.
- 348 doi:10.1016/j.injury.2017.08.040
- 349 33. Metsemakers WJ, Morgenstern M, McNally MA, et al. Fracture-related infection: A
- 350 consensus on definition from an international expert group. *Injury*. 2018;49:505-510.
- 351 34. Metsemakers WJ, Kuehl R, Moriarty TF, et al. Infection after fracture fixation: Current
- 352 surgical and microbiological concepts. *Injury*. 2018;49(3):511-522.
- 353 35. Study to Prospectively Evaluate Reamed Intramedullary Nails in Patients with Tibial
- 354 Fractures Investigators, Bhandari M, Guyatt G, et al. Randomized Trial of Reamed and
- 355 Unreamed Intramedullary Nailing of Tibial Shaft Fractures. J Bone Jt Surg-Am Vol.
- 356 2008;90(12):2567-2578.
- 357 36. Zampieri FG, Casey JD, Shankar-Hari M, Harrell FE, Harhay MO. Using Bayesian
- Methods to Augment the Interpretation of Critical Care Trials. An Overview of Theory and 358
- 359 Example Reanalysis of the Alveolar Recruitment for Acute Respiratory Distress Syndrome
- 360 Trial. Am J Respir Crit Care Med. 2021;203(5):543-552. doi:10.1164/rccm.202006-
- 361 2381CP